CLINICAL TRIAL: NCT02414854
Title: A Randomized, Double Blind, Placebo-Controlled, Parallel Group Study to Evaluate the Efficacy and Safety of Dupilumab in Patients With Persistent Asthma
Brief Title: Evaluation of Dupilumab in Patients With Persistent Asthma (Liberty Asthma Quest)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EFC13579; 2014-004940-36 (EudraCT Number); U1111-1163-1293 (Other: UTN)
Record Dates: First submitted 2015-04-08; First posted 2015-04-13 (Estimated); Results first posted 2018-10-23 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-06

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — dupilumab; Therapeutics; Albuterol; Levalbuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (for Dupilumab 200 mg) q2w (Placebo Comparator): 2 subcutaneous injections of matched Placebo (for Dupilumab 200 mg) as a loading dose on Day 1 (Week 0), followed by a single injection every 2 weeks (q2w) from Week 2 to Week 50 in combination with stable ICS and up to 2 other controller medicines. Albuterol/salbutamol or levalbuterol/levosalbutamol was given as reliever medication.
  Interventions: Drug: Placebo; Drug: Inhaled corticosteroid (ICS) therapy; Drug: Albuterol/Salbutamol; Drug: Levalbuterol/Levosalbutamol
- Dupilumab 200 mg q2w (Experimental): 2 subcutaneous injections of Dupilumab 200 mg (for a total of 400 mg) as a loading dose on Day 1 (Week 0), followed by a single 200 mg injection q2w from Week 2 to Week 50 in combination with stable ICS and up to 2 other controller medicines. Albuterol/salbutamol or levalbuterol/levosalbutamol was given as reliever medication.
  Interventions: Drug: Dupilumab; Drug: Inhaled corticosteroid (ICS) therapy; Drug: Albuterol/Salbutamol; Drug: Levalbuterol/Levosalbutamol
- Placebo (for Dupilumab 300 mg) q2w (Placebo Comparator): 2 subcutaneous injections of matched Placebo (for Dupilumab 300 mg) as a loading dose on Day 1 (Week 0), followed by a single injection q2w from Week 2 to Week 50 in combination with stable ICS and up to 2 other controller medicines. Albuterol/salbutamol or levalbuterol/levosalbutamol was given as reliever medication.
  Interventions: Drug: Placebo; Drug: Inhaled corticosteroid (ICS) therapy; Drug: Albuterol/Salbutamol; Drug: Levalbuterol/Levosalbutamol
- Dupilumab 300 mg q2w (Experimental): 2 subcutaneous injections of Dupilumab 300 mg (for a total of 600 mg) as a loading dose on Day 1 (Week 0), followed by a single 300 mg injection q2w from Week 2 to Week 50 in combination with stable ICS and up to 2 other controller medicines . Albuterol/salbutamol or levalbuterol/levosalbutamol was given as reliever medication.
  Interventions: Drug: Dupilumab; Drug: Inhaled corticosteroid (ICS) therapy; Drug: Albuterol/Salbutamol; Drug: Levalbuterol/Levosalbutamol

INTERVENTIONS:
Drug: Dupilumab — Solution for injection, Subcutaneous injection in the abdomen, upper thigh or upper arm.
  Other Names: SAR231893; REGN668
  Arms: Dupilumab 200 mg q2w; Dupilumab 300 mg q2w
Drug: Placebo — Solution for injection, Subcutaneous injection in the abdomen, upper thigh or upper arm.
  Arms: Placebo (for Dupilumab 200 mg) q2w; Placebo (for Dupilumab 300 mg) q2w
Drug: Inhaled corticosteroid (ICS) therapy — Oral inhalation, stable dose (medium or high dose) of ICS in combination with up to 2 other controller medicines (second or third controller therapy)
Drug: Albuterol/Salbutamol — Oral inhalation as needed
Drug: Levalbuterol/Levosalbutamol — Oral inhalation as needed

SUMMARY:
Primary Objective:

To evaluate the efficacy of dupilumab (SAR231893 / REGN668) in participants with persistent asthma.

Secondary Objectives:

* To evaluate the safety and tolerability of dupilumab.
* To evaluate the effect of dupilumab on improving participant-reported outcomes including health-related quality of life.
* To evaluate dupilumab systemic exposure and incidence of anti-drug antibodies.

DETAILED DESCRIPTION:
The total duration of study period for each participant is 67 to 69 weeks, including a screening period of 3 to 5 weeks, treatment period of 52 weeks, and post-treatment follow-up period of 12 weeks.

ELIGIBILITY:
Inclusion criteria:

-Adults and adolescent participants with a physician diagnosis of asthma for ≥12 months, based on the Global Initiative for Asthma (GINA) 2014 Guidelines and the following criteria:

a) Existing treatment with medium to high dose ICS (≥250 mcg of fluticasone propionate twice daily or equipotent ICS daily dosage to a maximum of 2000 mcg/day of fluticasone propionate or equivalent) in combination with a second controller (eg, long-acting beta agonist, leukotriene receptor antagonist) for at least 3 months with a stable dose ≥1 month prior to Visit 1.

i) Note for Japan: for participants aged 18 years and older, ICS must be on ≥200 mcg of fluticasone propionate twice daily or equivalent; for participants aged 12 to 17 years, ICS must be ≥100 mcg of fluticasone propionate twice daily or equivalent).

ii) Participants requiring a third controller for their asthma will be considered eligible for this study, and it should also be used for at least 3 months with a stable dose ≥1 month prior to Visit 1.

Exclusion criteria:

* Participants <12 years of age or the minimum legal age for adolescents in the country of the investigative site, whichever is higher (For those countries where local regulations permit enrollment of adults only, participant recruitment will be restricted to those who are ≥18 years of age).
* Weight is less than 30 kilograms.
* Chronic obstructive pulmonary disease or other lung diseases (eg, idiopathic pulmonary fibrosis, Churg-Strauss Syndrome, etc) which may impair lung function.
* A participant who experiences a severe asthma exacerbation (defined as a deterioration of asthma that results in emergency treatment, hospitalization due to asthma, or treatment with systemic steroids at any time from 1 month prior to the Screening Visit up to and including the Baseline Visit).
* Evidence of lung disease(s) other than asthma, either clinical evidence or imaging (Chest X-ray, CT, MRI) within 12 months of Visit 1 or at the screening visit, as per local standard of care.
* Note for Japan: According to the request from the health authority, chest X-ray should be performed at screening visit if there is no chest imaging (Chest X-ray, computed tomography [CT], magnetic resonance imaging [MRI]) available within 3 months prior to screening to exclude participants with suspected active or untreated latent tuberculosis.
* Current smoker or cessation of smoking within 6 months prior to Visit 1.
* Previous smoker with a smoking history >10 pack-years.
* Comorbid disease that might interfere with the evaluation of Investigational Medicinal Product.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1902 (Actual)
Dates: Start 2015-04-27; Primary Completion 2017-07-29 (Actual); Study Completion 2017-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (389):
- United States (116):
  - Investigational Site Number 840047, Birmingham, Alabama
  - Investigational Site Number 840056, Flagstaff, Arizona
  - Investigational Site Number 840099, Gilbert, Arizona
  - Investigational Site Number 840087, Scottsdale, Arizona
  - Investigational Site Number 840132, Little Rock, Arkansas
  - Investigational Site Number 840109, Bakersfield, California
  - Investigational Site Number 840052, Costa Mesa, California
  - Investigational Site Number 840116, Fresno, California
  - Investigational Site Number 840045, Long Beach, California
  - Investigational Site Number 840011, Los Angeles, California
  - Investigational Site Number 840061, Los Angeles, California
  - Investigational Site Number 840097, Los Angeles, California
  - Investigational Site Number 840019, Mission Viejo, California
  - Investigational Site Number 840125, Newport Beach, California
  - Investigational Site Number 840041, North Hollywood, California
  - Investigational Site Number 840036, Redwood City, California
  - Investigational Site Number 840020, Rolling Hills Estates, California
  - Investigational Site Number 840074, Roseville, California
  - Investigational Site Number 840021, San Jose, California
  - Investigational Site Number 840004, Centennial, Colorado
  - Investigational Site Number 840025, Colorado Springs, Colorado
  - Investigational Site Number 840034, Denver, Colorado
  - Investigational Site Number 840130, Denver, Colorado
  - Investigational Site Number 840102, New Haven, Connecticut
  - Investigational Site Number 840037, Aventura, Florida
  - Investigational Site Number 840018, Boynton Beach, Florida
  - Investigational Site Number 840105, Brandon, Florida
  - Investigational Site Number 840092, Clearwater, Florida
  - Investigational Site Number 840122, Hialeah, Florida
  - Investigational Site Number 840053, Loxahatchee Groves, Florida
  - Investigational Site Number 840069, Miami, Florida
  - Investigational Site Number 840123, Ocala, Florida
  - Investigational Site Number 840071, Ocala, Florida
  - Investigational Site Number 840115, Ocoee, Florida
  - Investigational Site Number 840055, Sarasota, Florida
  - Investigational Site Number 840114, South Miami, Florida
  - Investigational Site Number 840048, Tampa, Florida
  - Investigational Site Number 840084, Gainesville, Georgia
  - Investigational Site Number 840044, Savannah, Georgia
  - Investigational Site Number 840079, Twin Falls, Idaho
  - Investigational Site Number 840101, Chicago, Illinois
  - Investigational Site Number 840015, River Forest, Illinois
  - Investigational Site Number 840089, Iowa City, Iowa
  - Investigational Site Number 840032, Fort Mitchell, Kentucky
  - Investigational Site Number 840009, Owensboro, Kentucky
  - Investigational Site Number 840064, Bangor, Maine
  - Investigational Site Number 840080, Baltimore, Maryland
  - Investigational Site Number 840017, Chevy Chase, Maryland
  - Investigational Site Number 840073, Gaithersburg, Maryland
  - Investigational Site Number 840127, White Marsh, Maryland
  - Investigational Site Number 840014, North Dartmouth, Massachusetts
  - Investigational Site Number 840005, Minneapolis, Minnesota
  - Investigational Site Number 840013, Kansas City, Missouri
  - Investigational Site Number 840002, St Louis, Missouri
  - Investigational Site Number 840093, St Louis, Missouri
  - Investigational Site Number 840026, Missoula, Montana
  - Investigational Site Number 840078, Omaha, Nebraska
  - Investigational Site Number 840003, Papillion, Nebraska
  - Investigational Site Number 840111, Brick, New Jersey
  - Investigational Site Number 840068, Ocean City, New Jersey
  - Investigational Site Number 840016, Princeton, New Jersey
  - Investigational Site Number 840096, Toms River, New Jersey
  - Investigational Site Number 840106, Jamaica, New York
  - Investigational Site Number 840065, New York, New York
  - Investigational Site Number 840076, Rochester, New York
  - Investigational Site Number 840031, The Bronx, New York
  - Investigational Site Number 840126, Charlotte, North Carolina
  - Investigational Site Number 840083, Charlotte, North Carolina
  - Investigational Site Number 840108, Durham, North Carolina
  - Investigational Site Number 840107, Greensboro, North Carolina
  - Investigational Site Number 840007, High Point, North Carolina
  - Investigational Site Number 840046, Cincinnati, Ohio
  - Investigational Site Number 840049, Middleburg Heights, Ohio
  - Investigational Site Number 840042, Toledo, Ohio
  - Investigational Site Number 840112, Edmond, Oklahoma
  - Investigational Site Number 840121, Oklahoma City, Oklahoma
  - Investigational Site Number 840104, Tulsa, Oklahoma
  - Investigational Site Number 840040, Clackamas, Oregon
  - Investigational Site Number 840039, Medford, Oregon
  - Investigational Site Number 840001, Portland, Oregon
  - Investigational Site Number 840085, Hershey, Pennsylvania
  - Investigational Site Number 840081, Philadelphia, Pennsylvania
  - Investigational Site Number 840010, Philadelphia, Pennsylvania
  - Investigational Site Number 840067, Philadelphia, Pennsylvania
  - Investigational Site Number 840028, Pittsburgh, Pennsylvania
  - Investigational Site Number 840091, Pittsburgh, Pennsylvania
  - Investigational Site Number 840029, Lincoln, Rhode Island
  - Investigational Site Number 840082, Charleston, South Carolina
  - Investigational Site Number 840117, Greenville, South Carolina
  - Investigational Site Number 840100, Greer, South Carolina
  - Investigational Site Number 840054, Spartanburg, South Carolina
  - Investigational Site Number 840062, Amarillo, Texas
  - Investigational Site Number 840098, Austin, Texas
  - Investigational Site Number 840038, Boerne, Texas
  - Investigational Site Number 840124, Cypress, Texas
  - Investigational Site Number 840008, Dallas, Texas
  - Investigational Site Number 840094, Dallas, Texas
  - Investigational Site Number 840023, El Paso, Texas
  - Investigational Site Number 840022, Fort Worth, Texas
  - Investigational Site Number 840027, Fort Worth, Texas
  - Investigational Site Number 840066, Killeen, Texas
  - Investigational Site Number 840050, Live Oak, Texas
  - Investigational Site Number 840070, McKinney, Texas
  - Investigational Site Number 840128, McKinney, Texas
  - Investigational Site Number 840118, Plano, Texas
  - Investigational Site Number 840012, San Antonio, Texas
  - Investigational Site Number 840129, San Antonio, Texas
  - Investigational Site Number 840133, Sealy, Texas
  - Investigational Site Number 840119, Spring, Texas
  - Investigational Site Number 840035, Draper, Utah
  - Investigational Site Number 840077, Murray, Utah
  - Investigational Site Number 840057, South Burlington, Vermont
  - Investigational Site Number 840059, Fairfax, Virginia
  - Investigational Site Number 840113, Richmond, Virginia
  - Investigational Site Number 840051, Bellevue, Washington
  - Investigational Site Number 840043, Spokane, Washington
- Argentina (12):
  - Investigational Site Number 032006, Bahía Blanca
  - Investigational Site Number 032002, Buenos Aires
  - Investigational Site Number 032011, Caba
  - Investigational Site Number 032007, Caba
  - Investigational Site Number 032001, Caba
  - Investigational Site Number 032003, Caba
  - Investigational Site Number 032010, Caba
  - Investigational Site Number 032005, Capital Federal
  - Investigational Site Number 032008, La Plata
  - Investigational Site Number 032004, Rosario
  - Investigational Site Number 032012, San Miguel de Tucumán
  - Investigational Site Number 032009, San Miguel de Tucumán
- Australia (6):
  - Investigational Site Number 036005, Campbelltown
  - Investigational Site Number 036001, Clayton
  - Investigational Site Number 036002, Frankston
  - Investigational Site Number 036006, Glen Osmond
  - Investigational Site Number 036003, Murdoch
  - Investigational Site Number 036004, Parkville
- Brazil (9):
  - Investigational Site Number 076009, Florianópolis
  - Investigational Site Number 076007, Porto Alegre
  - Investigational Site Number 076001, Porto Alegre
  - Investigational Site Number 076003, Salvador
  - Investigational Site Number 076013, São Bernardo do Campo
  - Investigational Site Number 076012, São Paulo
  - Investigational Site Number 076008, São Paulo
  - Investigational Site Number 076006, São Paulo
  - Investigational Site Number 076002, Sorocaba
- Canada (14):
  - Investigational Site Number 124019, Burlington
  - Investigational Site Number 124009, Calgary
  - Investigational Site Number 124003, Mississauga
  - Investigational Site Number 124001, Montreal
  - Investigational Site Number 124012, Montreal
  - Investigational Site Number 124010, Montreal
  - Investigational Site Number 124013, Ottawa
  - Investigational Site Number 124018, Québec
  - Investigational Site Number 124014, Québec
  - Investigational Site Number 124008, Sherbrooke
  - Investigational Site Number 124015, Toronto
  - Investigational Site Number 124002, Toronto
  - Investigational Site Number 124007, Trois-Rivières
  - Investigational Site Number 124006, Vancouver
- Chile (16):
  - Investigational Site Number 152015, Concepción
  - Investigational Site Number 152003, Quillota
  - Investigational Site Number 152014, Santiago
  - Investigational Site Number 152001, Santiago
  - Investigational Site Number 152002, Santiago
  - Investigational Site Number 152008, Santiago
  - Investigational Site Number 152017, Santiago
  - Investigational Site Number 152007, Santiago
  - Investigational Site Number 152005, Santiago
  - Investigational Site Number 152009, Santiago
  - Investigational Site Number 152004, Talca
  - Investigational Site Number 152013, Talcahuano
  - Investigational Site Number 152016, Temuco
  - Investigational Site Number 152010, Valdivia
  - Investigational Site Number 152011, Viña del Mar
  - Investigational Site Number 152012, Viña del Mar
- Colombia (4):
  - Investigational Site Number 170006, Bogotá
  - Investigational Site Number 170001, Bogotá
  - Investigational Site Number 170002, Bogotá
  - Investigational Site Number 170003, Bogotá
- France (11):
  - Investigational Site Number 250002, Brest
  - Investigational Site Number 250013, Lille
  - Investigational Site Number 250011, Lille
  - Investigational Site Number 250004, Lyon
  - Investigational Site Number 250010, Marseille
  - Investigational Site Number 250005, Montpellier
  - Investigational Site Number 250003, Nantes
  - Investigational Site Number 250012, Paris
  - Investigational Site Number 250001, Paris
  - Investigational Site Number 250008, Strasbourg
  - Investigational Site Number 250014, Vandœuvre-lès-Nancy
- Germany (8):
  - Investigational Site Number 276006, Berlin
  - Investigational Site Number 276003, Bochum
  - Investigational Site Number 276010, Frankfurt am Main
  - Investigational Site Number 276004, Hanover
  - Investigational Site Number 276009, Koblenz
  - Investigational Site Number 276007, Lübeck
  - Investigational Site Number 276001, Mainz
  - Investigational Site Number 276005, Rüdersdorf
- Investigational Site Number 348003, Gödöllö, Hungary
- Italy (10):
  - Investigational Site Number 380004, Ancona
  - Investigational Site Number 380005, Catania
  - Investigational Site Number 380003, Ferrara
  - Investigational Site Number 380006, Florence
  - Investigational Site Number 380010, Foggia
  - Investigational Site Number 380002, Modena
  - Investigational Site Number 380009, Palermo
  - Investigational Site Number 380001, Pisa
  - Investigational Site Number 380014, Reggio Emilia
  - Investigational Site Number 380011, Torino
- Japan (72):
  - Investigational Site Number 392185, Akashi-Shi
  - Investigational Site Number 392128, Asahikawa-Shi
  - Investigational Site Number 392118, Chiyoda-Ku
  - Investigational Site Number 392112, Chūōku
  - Investigational Site Number 392157, Fukui-shi
  - Investigational Site Number 392137, Fukuoka
  - Investigational Site Number 392117, Fukuyama-Shi
  - Investigational Site Number 392121, Habikino-Shi
  - Investigational Site Number 392154, Higashiosaka-Shi
  - Investigational Site Number 392109, Himeji-Shi
  - Investigational Site Number 392108, Hiroshima
  - Investigational Site Number 392158, Hiroshima
  - Investigational Site Number 392107, Iizuka-Shi
  - Investigational Site Number 392101, Isesaki-Shi
  - Investigational Site Number 392147, Itabashi-Ku
  - Investigational Site Number 392150, Kagoshima
  - Investigational Site Number 392178, Kagoshima
  - Investigational Site Number 392110, Kanazawa
  - Investigational Site Number 392136, Kanazawa
  - Investigational Site Number 392142, Kasuga-Shi
  - Investigational Site Number 392166, Kawaguchi-Shi
  - Investigational Site Number 392119, Kishiwada-Shi
  - Investigational Site Number 392162, Kobe
  - Investigational Site Number 392182, Kodaira-Shi
  - Investigational Site Number 392174, Kokubunji-Shi
  - Investigational Site Number 392131, Koshi-Shi
  - Investigational Site Number 392183, Koshigaya-Shi
  - Investigational Site Number 392129, Kurashiki-Shi
  - Investigational Site Number 392153, Kyoto
  - Investigational Site Number 392176, Kyoto
  - Investigational Site Number 392184, Kyoto
  - Investigational Site Number 392133, Machida-Shi
  - Investigational Site Number 392135, Matsuyama
  - Investigational Site Number 392172, Mibu
  - Investigational Site Number 392114, Minatoku
  - Investigational Site Number 392122, Minatoku
  - Investigational Site Number 392144, Minatoku
  - Investigational Site Number 392106, Mizunami-Shi
  - Investigational Site Number 392164, Muroran-Shi
  - Investigational Site Number 392161, Nagakute-Shi
  - Investigational Site Number 392163, Nagoya
  - Investigational Site Number 392102, Naka-Gun
  - Investigational Site Number 392125, Nakano
  - Investigational Site Number 392115, Naruto-Shi
  - Investigational Site Number 392187, Obihiro-Shi
  - Investigational Site Number 392177, Ome-Shi
  - Investigational Site Number 392152, Osaka Sayama-Shi
  - Investigational Site Number 392155, Osaka Sayama-Shi
  - Investigational Site Number 392170, Osaki-Shi
  - Investigational Site Number 392138, Ota-Shi
  - Investigational Site Number 392123, Oura-Gun
  - Investigational Site Number 392120, Ōta-ku
  - Investigational Site Number 392127, Ōta-ku
  - Investigational Site Number 392169, Sagamihara-Shi
  - Investigational Site Number 392149, Sapporo
  - Investigational Site Number 392179, Seto-Shi
  - Investigational Site Number 392186, Shibuya-Ku
  - Investigational Site Number 392139, Shinagawa-Ku
  - Investigational Site Number 392167, Shinagawa-Ku
  - Investigational Site Number 392130, Shinjuku-Ku
  - Investigational Site Number 392165, Sumida-Ku
  - Investigational Site Number 392146, Tachikawa-Shi
  - Investigational Site Number 392173, Tachikawa-Shi
  - Investigational Site Number 392103, Tokyo
  - Investigational Site Number 392113, Tomakomai-Shi
  - Investigational Site Number 392151, Tsu
  - Investigational Site Number 392168, Uozu-Shi
  - Investigational Site Number 392132, Urasoe-Shi
  - Investigational Site Number 392134, Uruma
  - Investigational Site Number 392116, Wakayama
  - Investigational Site Number 392140, Yokohama
  - Investigational Site Number 392159, Yonago-Shi
- Mexico (12):
  - Investigational Site Number 484013, Chihuahua City
  - Investigational Site Number 484006, Chihuahua City
  - Investigational Site Number 484014, Cuautitlán Izcalli
  - Investigational Site Number 484008, Durango
  - Investigational Site Number 484001, Guadalajara
  - Investigational Site Number 484004, Mexico City
  - Investigational Site Number 484010, México
  - Investigational Site Number 484003, Monterrey
  - Investigational Site Number 484007, Monterrey
  - Investigational Site Number 484012, San Juan del Río
  - Investigational Site Number 484011, Veracruz
  - Investigational Site Number 484015, Zapopan
- Poland (9):
  - Investigational Site Number 616006, Bialystok
  - Investigational Site Number 616003, Gdansk
  - Investigational Site Number 616007, Krakow
  - Investigational Site Number 616001, Lodz
  - Investigational Site Number 616005, Lodz
  - Investigational Site Number 616009, Lodz
  - Investigational Site Number 616002, Poznan
  - Investigational Site Number 616004, Sopot
  - Investigational Site Number 616008, Strzelce Opolskie
- Russia (13):
  - Investigational Site Number 643006, Moscow
  - Investigational Site Number 643003, Moscow
  - Investigational Site Number 643005, Moscow
  - Investigational Site Number 643002, Moscow
  - Investigational Site Number 643004, Moscow
  - Investigational Site Number 643001, Moscow
  - Investigational Site Number 643011, Ryazan
  - Investigational Site Number 643007, Saint Petersburg
  - Investigational Site Number 643008, Saint Petersburg
  - Investigational Site Number 643009, Saint Petersburg
  - Investigational Site Number 643010, Saint Petersburg
  - Investigational Site Number 643012, Yaroslavl
  - Investigational Site Number 643013, Yekaterinburg
- South Africa (10):
  - Investigational Site Number 710011, Cape Town
  - Investigational Site Number 710004, Cape Town
  - Investigational Site Number 710001, Cape Town
  - Investigational Site Number 710002, Cape Town
  - Investigational Site Number 710010, Cape Town
  - Investigational Site Number 710003, Cape Town
  - Investigational Site Number 710005, Durban
  - Investigational Site Number 710006, Durban
  - Investigational Site Number 710007, Pretoria
  - Investigational Site Number 710009, Winnie Mandela
- South Korea (15):
  - Investigational Site Number 410002, Bucheon-si
  - Investigational Site Number 410015, Busan
  - Investigational Site Number 410003, Cheongju-si
  - Investigational Site Number 410013, Incheon
  - Investigational Site Number 410008, Seoul
  - Investigational Site Number 410006, Seoul
  - Investigational Site Number 410004, Seoul
  - Investigational Site Number 410012, Seoul
  - Investigational Site Number 410005, Seoul
  - Investigational Site Number 410007, Seoul
  - Investigational Site Number 410009, Seoul
  - Investigational Site Number 410010, Seoul
  - Investigational Site Number 410011, Seoul
  - Investigational Site Number 410001, Suwon
  - Investigational Site Number 410014, Uijeongbu-si
- Spain (8):
  - Investigational Site Number 724002, Barcelona
  - Investigational Site Number 724001, Barcelona
  - Investigational Site Number 724010, Palma de Mallorca
  - Investigational Site Number 724005, Pozuelo de Alarcón
  - Investigational Site Number 724004, Sant Boi de Llobregat
  - Investigational Site Number 724006, Santiago de Compostela
  - Investigational Site Number 724008, Seville
  - Investigational Site Number 724007, Valencia
- Taiwan (8):
  - Investigational Site Number 158004, Kaohsiung City
  - Investigational Site Number 158002, Kaohsiung City
  - Investigational Site Number 158008, New Taipei City
  - Investigational Site Number 158005, Taichung
  - Investigational Site Number 158007, Taichung
  - Investigational Site Number 158001, Taipei
  - Investigational Site Number 158009, Taipei
  - Investigational Site Number 158006, Taoyuan District
- Turkey (Türkiye) (11):
  - Investigational Site Number 792004, Ankara
  - Investigational Site Number 792008, Ankara
  - Investigational Site Number 792003, Bursa
  - Investigational Site Number 792001, Istanbul
  - Investigational Site Number 792007, Istanbul
  - Investigational Site Number 792005, Izmir
  - Investigational Site Number 792010, Izmir
  - Investigational Site Number 792011, Kocaeli
  - Investigational Site Number 792009, Kırıkkale
  - Investigational Site Number 792002, Mersin
  - Investigational Site Number 792006, Rize
- Ukraine (18):
  - Investigational Site Number 804007, Chernivtsi
  - Investigational Site Number 804023, Dnipro
  - Investigational Site Number 804004, Ivano-Frankivsk
  - Investigational Site Number 804009, Ivano-Frankivsk
  - Investigational Site Number 804005, Kharkiv
  - Investigational Site Number 804021, Kharkiv
  - Investigational Site Number 804001, Kharkiv
  - Investigational Site Number 804003, Kyiv
  - Investigational Site Number 804008, Kyiv
  - Investigational Site Number 804011, Kyiv
  - Investigational Site Number 804013, Kyiv
  - Investigational Site Number 804017, Kyiv
  - Investigational Site Number 804016, Kyiv
  - Investigational Site Number 804006, Odesa
  - Investigational Site Number 804002, Poltava
  - Investigational Site Number 804014, Ternopil
  - Investigational Site Number 804012, Vinnytsia
  - Investigational Site Number 804022, Zaporizhia
- United Kingdom (6):
  - Investigational Site Number 826001, Bradford
  - Investigational Site Number 826002, London
  - Investigational Site Number 826005, Newcastle upon Tyne
  - Investigational Site Number 826007, Portsmouth
  - Investigational Site Number 826006, South Shields
  - Investigational Site Number 826003, Sutton in Ashfield

REFERENCES:
- [Result] Castro M, Corren J, Pavord ID, Maspero J, Wenzel S, Rabe KF, Busse WW, Ford L, Sher L, FitzGerald JM, Katelaris C, Tohda Y, Zhang B, Staudinger H, Pirozzi G, Amin N, Ruddy M, Akinlade B, Khan A, Chao J, Martincova R, Graham NMH, Hamilton JD, Swanson BN, Stahl N, Yancopoulos GD, Teper A. Dupilumab Efficacy and Safety in Moderate-to-Severe Uncontrolled Asthma. N Engl J Med. 2018 Jun 28;378(26):2486-2496. doi: 10.1056/NEJMoa1804092. Epub 2018 May 21. PMID 29782217
- [Derived] Pavord ID, Wechsler ME, Busse WW, Domingo C, Xia C, Gall R, Pandit-Abid N, Jacob-Nara JA, Radwan A, Rowe PJ, Deniz Y. Dupilumab efficacy in patients with type 2 asthma and early Feno level reductions. J Allergy Clin Immunol Glob. 2025 Apr 15;4(3):100474. doi: 10.1016/j.jacig.2025.100474. eCollection 2025 Aug. PMID 40458676
- [Derived] Pavord ID, Casale TB, Corren J, FitzGerald MJ, Deniz Y, Altincatal A, Gall R, Pandit-Abid N, Radwan A, Jacob-Nara JA, Rowe PJ, Busse WW. Dupilumab Reduces Exacerbations Independent of Changes in Biomarkers in Moderate-to-Severe Asthma. J Allergy Clin Immunol Pract. 2024 Jul;12(7):1763-1772. doi: 10.1016/j.jaip.2024.03.031. Epub 2024 Mar 29. PMID 38555079
- [Derived] Peters AT, Sagara H, Corren J, Domingo C, Altincatal A, Soler X, Pandit-Abid N, Crikelair N, Rowe PJ, Jacob-Nara JA, Deniz Y. Impact of dupilumab across seasons in patients with type 2, uncontrolled, moderate-to-severe asthma. Ann Allergy Asthma Immunol. 2024 Apr;132(4):477-484.e4. doi: 10.1016/j.anai.2023.11.021. Epub 2023 Nov 25. PMID 38013139
- [Derived] Bleecker ER, Panettieri RA Jr, Lugogo NL, Corren J, Daizadeh N, Jacob-Nara JA, Deniz Y, Rowe PJ, Khodzhayev A, Soler X, Ferro TJ, Hansen CN. Dupilumab Efficacy in Patients with Type 2 Asthma with and without Elevated Blood Neutrophils. J Immunol Res. 2023 Oct 19;2023:9943584. doi: 10.1155/2023/9943584. eCollection 2023. PMID 37901346
- [Derived] Corren J, Hanania NA, Busse WW, Sher LD, Altincatal A, Hardin M, Mannent LP, Amin N, Lederer DJ, Soler X, Jacob-Nara JA, Rowe PJ, Deniz Y. Efficacy of dupilumab in patients with uncontrolled, moderate-to-severe asthma with fungal sensitization. Clin Exp Allergy. 2023 Oct;53(10):1020-1030. doi: 10.1111/cea.14389. Epub 2023 Sep 26. PMID 37752621
- [Derived] Maspero JF, Shafazand S, Cole J, Pavord ID, Busse WW, Msihid J, Gall R, Soler X, Radwan A, Khan AH, de Prado Gomez L, Jacob-Nara JA. Dupilumab efficacy in high sleep disturbance management among patients with type 2 asthma. Respir Med. 2023 Nov;218:107344. doi: 10.1016/j.rmed.2023.107344. Epub 2023 Sep 1. PMID 37659435
- [Derived] Pavord ID, Bourdin A, Papi A, Domingo C, Corren J, Altincatal A, Radwan A, Pandit-Abid N, Jacob-Nara JA, Deniz Y, Rowe PJ, Laws E, Lederer DJ, Hardin M. Dupilumab sustains efficacy in patients with moderate-to-severe type 2 asthma regardless of inhaled corticosteroids dose. Allergy. 2023 Nov;78(11):2921-2932. doi: 10.1111/all.15792. Epub 2023 Jul 11. PMID 37431558
- [Derived] Rabe KF, Pavord ID, Busse WW, Chupp GL, Izuhara K, Altincatal A, Gall R, Pandit-Abid N, Deniz Y, Rowe PJ, Jacob-Nara JA, Radwan A. Dupilumab improves long-term outcomes in patients with uncontrolled, moderate-to-severe GINA-based type 2 asthma, irrespective of allergic status. Allergy. 2023 Aug;78(8):2148-2156. doi: 10.1111/all.15747. Epub 2023 May 21. PMID 37073882
- [Derived] Pavord ID, Deniz Y, Corren J, Casale TB, FitzGerald JM, Izuhara K, Daizadeh N, Ortiz B, Johnson RR, Harel S, Djandji M, Goga L, Crikelair N, Rowe PJ, Busse WW. Baseline FeNO Independently Predicts the Dupilumab Response in Patients With Moderate-to-Severe Asthma. J Allergy Clin Immunol Pract. 2023 Apr;11(4):1213-1220.e2. doi: 10.1016/j.jaip.2022.11.043. Epub 2022 Dec 16. PMID 36535524
- [Derived] Berger P, Menzies-Gow A, Peters AT, Kuna P, Rabe KF, Altincatal A, Soler X, Pandit-Abid N, Siddiqui S, Jacob-Nara JA, Deniz Y, Rowe PJ. Long-term efficacy of dupilumab in asthma with or without chronic rhinosinusitis and nasal polyps. Ann Allergy Asthma Immunol. 2023 Feb;130(2):215-224. doi: 10.1016/j.anai.2022.11.006. Epub 2022 Nov 7. PMID 36356712
- [Derived] Bourdin A, Virchow JC, Papi A, Lugogo NL, Bardin P, Antila M, Halpin DMG, Daizadeh N, Djandji M, Ortiz B, Jacob-Nara JA, Gall R, Deniz Y, Rowe PJ. Dupilumab efficacy in subgroups of type 2 asthma with high-dose inhaled corticosteroids at baseline. Respir Med. 2022 Oct;202:106938. doi: 10.1016/j.rmed.2022.106938. Epub 2022 Aug 11. PMID 36087550
- [Derived] Rabe KF, FitzGerald JM, Bateman ED, Castro M, Pavord ID, Maspero JF, Busse WW, Izuhara K, Daizadeh N, Ortiz B, Pandit-Abid N, Rowe PJ, Deniz Y. Dupilumab Is Effective in Patients With Moderate-to-Severe Uncontrolled GINA-Defined Type 2 Asthma Irrespective of an Allergic Asthma Phenotype. J Allergy Clin Immunol Pract. 2022 Nov;10(11):2916-2924.e4. doi: 10.1016/j.jaip.2022.06.036. Epub 2022 Aug 23. PMID 36028446
- [Derived] Papi A, Corren J, Castro M, Domingo C, Rogers L, Chapman KR, Jackson DJ, Daizadeh N, Pandit-Abid N, Gall R, Jacob-Nara JA, Rowe PJ, Deniz Y, Ortiz B. Dupilumab reduced impact of severe exacerbations on lung function in patients with moderate-to-severe type 2 asthma. Allergy. 2023 Jan;78(1):233-243. doi: 10.1111/all.15456. Epub 2022 Aug 9. PMID 35899469
- [Derived] Wechsler ME, Klion AD, Paggiaro P, Nair P, Staumont-Salle D, Radwan A, Johnson RR, Kapoor U, Khokhar FA, Daizadeh N, Chen Z, Laws E, Ortiz B, Jacob-Nara JA, Mannent LP, Rowe PJ, Deniz Y. Effect of Dupilumab on Blood Eosinophil Counts in Patients With Asthma, Chronic Rhinosinusitis With Nasal Polyps, Atopic Dermatitis, or Eosinophilic Esophagitis. J Allergy Clin Immunol Pract. 2022 Oct;10(10):2695-2709. doi: 10.1016/j.jaip.2022.05.019. Epub 2022 May 28. PMID 35636689
- [Derived] Rabe KF, Pavord ID, Castro M, Wechsler ME, Daizadeh N, Kapoor U, Ortiz B, Radwan A, Johnson RR, Rowe PJ, Deniz Y, Jacob-Nara JA. Dupilumab efficacy and safety in patients with asthma and blood eosinophils >/=500 cells.microL-1. Eur Respir J. 2022 Jun 23;59(6):2102577. doi: 10.1183/13993003.02577-2021. Print 2022 Jun. PMID 35487538
- [Derived] Rhee CK, Park JW, Park HW, Cho YS. Effect of Dupilumab in Korean Patients With Uncontrolled Moderate-to-Severe Asthma: A LIBERTY ASTHMA QUEST Sub-analysis. Allergy Asthma Immunol Res. 2022 Mar;14(2):182-195. doi: 10.4168/aair.2022.14.2.182. PMID 35255536
- [Derived] Geng B, Bachert C, Busse WW, Gevaert P, Lee SE, Niederman MS, Chen Z, Lu X, Khokhar FA, Kapoor U, Pandit-Abid N, Jacob-Nara JA, Rowe PJ, Deniz Y, Ortiz B. Respiratory Infections and Anti-Infective Medication Use From Phase 3 Dupilumab Respiratory Studies. J Allergy Clin Immunol Pract. 2022 Mar;10(3):732-741. doi: 10.1016/j.jaip.2021.12.006. Epub 2021 Dec 22. PMID 34954123
- [Derived] Tohda Y, Matsumoto H, Miyata M, Taguchi Y, Ueyama M, Joulain F, Arakawa I. Cost-effectiveness analysis of dupilumab among patients with oral corticosteroid-dependent uncontrolled severe asthma in Japan. J Asthma. 2022 Nov;59(11):2162-2173. doi: 10.1080/02770903.2021.1996596. Epub 2021 Dec 8. PMID 34752208
- [Derived] Busse WW, Paggiaro P, Munoz X, Casale TB, Castro M, Canonica GW, Douglass JA, Tohda Y, Daizadeh N, Ortiz B, Pandit-Abid N. Impact of baseline patient characteristics on dupilumab efficacy in type 2 asthma. Eur Respir J. 2021 Oct 7;58(4):2004605. doi: 10.1183/13993003.04605-2020. Print 2021 Oct. PMID 34326187
- [Derived] Corren J, Katelaris CH, Castro M, Maspero JF, Ford LB, Halpin DMG, Rice MS, Radwan A, Deniz Y, Rowe PJ, Teper A, Djandji M. Effect of exacerbation history on clinical response to dupilumab in moderate-to-severe uncontrolled asthma. Eur Respir J. 2021 Oct 28;58(4):2004498. doi: 10.1183/13993003.04498-2020. Print 2021 Oct. PMID 34266940
- [Derived] Busse WW, Wenzel SE, Casale TB, FitzGerald JM, Rice MS, Daizadeh N, Deniz Y, Patel N, Harel S, Rowe PJ, Graham NMH, O'Riordan T, Pavord ID. Baseline FeNO as a prognostic biomarker for subsequent severe asthma exacerbations in patients with uncontrolled, moderate-to-severe asthma receiving placebo in the LIBERTY ASTHMA QUEST study: a post-hoc analysis. Lancet Respir Med. 2021 Oct;9(10):1165-1173. doi: 10.1016/S2213-2600(21)00124-7. Epub 2021 Jun 25. PMID 34181876
- [Derived] Hamilton JD, Harel S, Swanson BN, Brian W, Chen Z, Rice MS, Amin N, Ardeleanu M, Radin A, Shumel B, Ruddy M, Patel N, Pirozzi G, Mannent L, Graham NMH. Dupilumab suppresses type 2 inflammatory biomarkers across multiple atopic, allergic diseases. Clin Exp Allergy. 2021 Jul;51(7):915-931. doi: 10.1111/cea.13954. Epub 2021 Jun 26. PMID 34037993
- [Derived] Maspero JF, FitzGerald JM, Pavord ID, Rice MS, Maroni J, Rowe PJ, Pirozzi G, Amin N, Ruddy M, Graham NMH, Teper A, Hardin M. Dupilumab efficacy in adolescents with uncontrolled, moderate-to-severe asthma: LIBERTY ASTHMA QUEST. Allergy. 2021 Aug;76(8):2621-2624. doi: 10.1111/all.14872. Epub 2021 May 10. No abstract available. PMID 33905544
- [Derived] Bansal A, Simpson EL, Paller AS, Siegfried EC, Blauvelt A, de Bruin-Weller M, Corren J, Sher L, Guttman-Yassky E, Chen Z, Daizadeh N, Kamal MA, Shumel B, Mina-Osorio P, Mannent L, Patel N, Graham NMH, Khokhar FA, Ardeleanu M. Conjunctivitis in Dupilumab Clinical Trials for Adolescents with Atopic Dermatitis or Asthma. Am J Clin Dermatol. 2021 Jan;22(1):101-115. doi: 10.1007/s40257-020-00577-1. PMID 33481203
- [Derived] Bourdin A, Papi AA, Corren J, Virchow JC, Rice MS, Deniz Y, Djandji M, Rowe P, Pavord ID. Dupilumab is effective in type 2-high asthma patients receiving high-dose inhaled corticosteroids at baseline. Allergy. 2021 Jan;76(1):269-280. doi: 10.1111/all.14611. Epub 2020 Oct 21. PMID 33010038
- [Derived] Tohda Y, Nakamura Y, Fujisawa T, Ebisawa M, Arima K, Miyata M, Takahashi Y, Rice MS, Deniz Y, Rowe P, Patel N, Graham NMH, Teper A. Dupilumab efficacy and safety in Japanese patients with uncontrolled, moderate-to-severe asthma in the phase 3 LIBERTY ASTHMA QUEST study. Allergol Int. 2020 Oct;69(4):578-587. doi: 10.1016/j.alit.2020.04.002. Epub 2020 May 20. PMID 32444306
- [Derived] Corren J, Castro M, O'Riordan T, Hanania NA, Pavord ID, Quirce S, Chipps BE, Wenzel SE, Thangavelu K, Rice MS, Harel S, Jagerschmidt A, Khan AH, Kamat S, Maroni J, Rowe P, Lu Y, Amin N, Pirozzi G, Ruddy M, Graham NMH, Teper A. Dupilumab Efficacy in Patients with Uncontrolled, Moderate-to-Severe Allergic Asthma. J Allergy Clin Immunol Pract. 2020 Feb;8(2):516-526. doi: 10.1016/j.jaip.2019.08.050. Epub 2019 Sep 12. PMID 31521831
- [Derived] Maspero JF, Katelaris CH, Busse WW, Castro M, Corren J, Chipps BE, Peters AT, Pavord ID, Ford LB, Sher L, Rabe KF, Rice MS, Rowe P, Lu Y, Harel S, Jagerschmidt A, Khan AH, Kamat S, Pirozzi G, Amin N, Ruddy M, Graham NMH, Mannent LP, Teper A. Dupilumab Efficacy in Uncontrolled, Moderate-to-Severe Asthma with Self-Reported Chronic Rhinosinusitis. J Allergy Clin Immunol Pract. 2020 Feb;8(2):527-539.e9. doi: 10.1016/j.jaip.2019.07.016. Epub 2019 Jul 24. PMID 31351189
- [Derived] Corren J, Castro M, Chanez P, Fabbri L, Joish VN, Amin N, Graham NMH, Mastey V, Abbe A, Taniou C, Mahajan P, Teper A, Pirozzi G, Eckert L. Dupilumab improves symptoms, quality of life, and productivity in uncontrolled persistent asthma. Ann Allergy Asthma Immunol. 2019 Jan;122(1):41-49.e2. doi: 10.1016/j.anai.2018.08.005. Epub 2018 Aug 21. PMID 30138668
- [Derived] Busse WW, Maspero JF, Rabe KF, Papi A, Wenzel SE, Ford LB, Pavord ID, Zhang B, Staudinger H, Pirozzi G, Amin N, Akinlade B, Eckert L, Chao J, Graham NMH, Teper A. Liberty Asthma QUEST: Phase 3 Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate Dupilumab Efficacy/Safety in Patients with Uncontrolled, Moderate-to-Severe Asthma. Adv Ther. 2018 May;35(5):737-748. doi: 10.1007/s12325-018-0702-4. Epub 2018 May 3. PMID 29725983
- [Derived] Weinstein SF, Katial R, Jayawardena S, Pirozzi G, Staudinger H, Eckert L, Joish VN, Amin N, Maroni J, Rowe P, Graham NMH, Teper A. Efficacy and safety of dupilumab in perennial allergic rhinitis and comorbid asthma. J Allergy Clin Immunol. 2018 Jul;142(1):171-177.e1. doi: 10.1016/j.jaci.2017.11.051. Epub 2018 Jan 31. PMID 29355679
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/?term=29782217&report=abstract

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 4148 participants were screened from Apr 2015-Sep 2016. 1902 were randomized at 321 centers/22 countries. 2246 were screen failures. 1897 participants were treated; some received a different treatment than that assigned at randomization and for adverse event (AE) analysis were allocated to treatment actually received (see footnotes in below table)
Pre-assignment Details: Randomization was stratified by age (<18 years, >=18 years), blood eosinophil count(<0.3 Giga/L, >=0.3 Giga/L), ICS dose level (medium, high), and country. Assignment to arms was done centrally using Interactive Voice/Web Response System in 2:2:1:1 ratio to Dupilumab 200 mg q2w, Dupilumab 300 mg q2w, Placebo (for 200 mg)q2w, Placebo (for 300 mg)q2w
Groups:
- Placebo (for Dupilumab 200 mg) q2w: 2 subcutaneous injections of matched Placebo (for Dupilumab 200 mg) as a loading dose on Day 1 (Week 0), followed by a single injection every 2 weeks (q2w) from Week 2 to Week 50 in combination with stable inhaled corticosteroid (ICS) and up to 2 other controller medicines (second or third controller therapy). Albuterol/salbutamol or levalbuterol/levosalbutamol was given as reliever medication.
- Dupilumab 200 mg q2w: 2 subcutaneous injections of Dupilumab 200 mg (for a total of 400 mg) as a loading dose on Day 1 (Week 0), followed by a single 200 mg injection q2w from Week 2 to Week 50 in combination with stable ICS and up to 2 other controller medicines (second or third controller therapy). Albuterol/salbutamol or levalbuterol/levosalbutamol was given as reliever medication.
- Placebo (for Dupilumab 300 mg) q2w: 2 subcutaneous injections of matched Placebo (for Dupilumab 300 mg) as a loading dose on Day 1 (Week 0), followed by a single injection q2w from Week 2 to Week 50 in combination with stable ICS and up to 2 other controller medicines (second or third controller therapy). Albuterol/salbutamol or levalbuterol/levosalbutamol was given as reliever medication.
- Dupilumab 300 mg q2w: 2 subcutaneous injections of Dupilumab 300 mg (for a total of 600 mg) as a loading dose on Day 1 (Week 0), followed by a single 300 mg injection q2w from Week 2 to Week 50 in combination with stable ICS and up to 2 other controller medicines (second or third controller therapy). Albuterol/salbutamol or levalbuterol/levosalbutamol was given as reliever medication.
Period: Overall Study
Arm/Group | Placebo (for Dupilumab 200 mg) q2w | Dupilumab 200 mg q2w | Placebo (for Dupilumab 300 mg) q2w | Dupilumab 300 mg q2w
Started (Randomized) | 317 | 631 | 321 | 633
Treated (Randomized) | 315 (2 got other treatment (1 each dupilumab 200+300) than assigned + were allocated to those in AE table) | 629 | 321 | 632 (1 got other treatment (dupilumab 200) than assigned + was allocated to that in AE table)
Completed | 295 | 586 | 301 | 582
Not Completed | 22 | 45 | 20 | 51
Not completed — Adverse Event | 9 | 7 | 1 | 12
Not completed — Poor compliance to protocol | 1 | 1 | 2 | 2
Not completed — Other than specified above | 12 | 37 | 17 | 37

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all randomized participants.
Groups:
- Placebo (for Dupilumab 200 mg) q2w: 2 subcutaneous injections of matched Placebo (for Dupilumab 200 mg) as a loading dose on Day 1 (Week 0), followed by a single injection q2w from Week 2 to Week 50 in combination with stable ICS and up to 2 other controller medicines (second or third controller therapy). Albuterol/salbutamol or levalbuterol/levosalbutamol was given as reliever medication.
- Total: Total of all reporting groups
Arm/Group | Placebo (for Dupilumab 200 mg) q2w | Dupilumab 200 mg q2w | Placebo (for Dupilumab 300 mg) q2w | Dupilumab 300 mg q2w | Total
Number analyzed (Participants) | 317 | 631 | 321 | 633 | 1902
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.2 (15.6) | 47.9 (15.3) | 48.2 (14.7) | 47.7 (15.6) | 47.9 (15.3)
Age, Customized [Count of Participants; unit: Participants]
  Adolescents (12-17 years) | 21 | 34 | 18 | 34 | 107
  Adults (18-64 years) | 253 | 512 | 263 | 516 | 1544
  From 65-84 years | 43 | 85 | 40 | 83 | 251
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 198 | 387 | 218 | 394 | 1197
  Male | 119 | 244 | 103 | 239 | 705
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 81 | 171 | 79 | 159 | 490
  Not Hispanic or Latino | 236 | 460 | 242 | 474 | 1412
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian/White | 265 | 510 | 273 | 529 | 1577
  Black/of African descent | 14 | 33 | 12 | 21 | 80
  Asian/Oriental | 33 | 78 | 33 | 79 | 223
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  Other | 4 | 9 | 3 | 4 | 20
Blood Eosinophil Group [Count of Participants; unit: Participants] — Population: Number analyzed = Number of participants with eosinophil data.
  Participants
    <0.15 Giga/L: number analyzed (Participants) | 317 | 630 | 320 | 633 | 1900
    <0.15 Giga/L | 85 | 193 | 83 | 181 | 542
    >=0.15 - <0.3 Giga/L: number analyzed (Participants) | 317 | 630 | 320 | 633 | 1900
    >=0.15 - <0.3 Giga/L | 84 | 173 | 95 | 175 | 527
    >=0.3 Giga/L: number analyzed (Participants) | 317 | 630 | 320 | 633 | 1900
    >=0.3 Giga/L | 148 | 264 | 142 | 277 | 831
ICS Dose Level [Count of Participants; unit: Participants]
  High | 172 | 317 | 167 | 323 | 979
  Medium | 144 | 310 | 151 | 303 | 908
  Low | 1 | 4 | 3 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Annualized Rate of Severe Exacerbation Events During The 52-Week Treatment Period: Intent-to-Treat (ITT) Population
Description: A severe exacerbation was defined as a deterioration of asthma requiring: use of systemic corticosteroids for >=3 days; or hospitalization or emergency room visit because of asthma, requiring systemic corticosteroids. Annualized event rate was the total number of exacerbations that occurred during the treatment period divided by the total number of participant-years treated.
Time Frame: Baseline to Week 52
Population: Analysis was performed on ITT population that included all randomized population analyzed according to the treatment group allocated by randomization.
Measure: Number (95% Confidence Interval); unit: Exacerbation per participant-year
Arm/Group | Placebo (for Dupilumab 200 mg) q2w | Dupilumab 200 mg q2w | Placebo (for Dupilumab 300 mg) q2w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 317 | 631 | 321 | 633
Exacerbation per participant-year | 0.871 [0.724 to 1.048] | 0.456 [0.389 to 0.534] | 0.970 [0.810 to 1.160] | 0.524 [0.450 to 0.611]
Statistical Analysis 1: Comparison: Placebo (for Dupilumab 300 mg) q2w vs Dupilumab 300 mg q2w; Analysis was performed using negative binomial model with total number of events onset from randomization up to Week 52 or last contact date (whichever comes earlier) as response variable; with 4 treatment groups, age, region, baseline eosinophil strata, baseline ICS dose level, number of severe exacerbation events within 1 year prior to study as covariates; and log transformed standardized observation duration as an offset variable. Here, it is test no. 1 of testing order; Test type: Superiority — Hierarchical testing procedure was used to control type I error rate at 0.05 level. The procedure included the 2 primary outcome measures and the first 13 secondary outcome measures reported and considered 2 pair-wise comparisons: Dupilumab 200 mg q2w vs Placebo (for Dupilumab 200 mg) q2w and Dupilumab 300 mg q2w vs Placebo (for Dupilumab 300 mg) q2w. Testing order is specified in analysis description; p < 0.0001, Negative binomial regression model — Hierarchical testing sequence performed continued only when previous outcome measures was statistically significant at 0.05. Threshold for significance at 0.05 level; Relative risk = 0.54, 95% CI 2-sided [0.43 to 0.68] — Dupilumab 300 mg q2w vs Placebo (for Dupilumab 300 mg) q2w
Statistical Analysis 2: Comparison: Placebo (for Dupilumab 200 mg) q2w vs Dupilumab 200 mg q2w; Analysis was performed using negative binomial model with total number of events onset from randomization up to Week 52 or last contact date (whichever comes earlier) as response variable; with 4 treatment groups, age, region, baseline eosinophil strata, baseline ICS dose level, number of severe exacerbation events within 1 year prior to study as covariates; and log transformed standardized observation duration as an offset variable. Here, it is test no. 3 of testing order; Test type: Superiority — Testing according to the hierarchical testing procedure (performed only if previous outcome measures were statistically significant); p < 0.0001, Negative binomial regression model — Threshold for significance at 0.05 level; Relative risk = 0.523, 95% CI 2-sided [0.413 to 0.662] — Dupilumab 200 mg q2w vs Placebo (for Dupilumab 200 mg) q2w

2. Primary Outcome: Absolute Change From Baseline in Pre-Bronchodilator Forced Expiratory Volume in 1 Second (FEV1) at Week 12: ITT Population
Description: FEV1 was the volume of air exhaled in the first second of a forced expiration as measured by spirometer.
Time Frame: Baseline, Week 12
Population: Analysis was performed on ITT population. Here 'Number analyzed' signifies number of participants with available data for specified category.
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | Placebo (for Dupilumab 200 mg) q2w | Dupilumab 200 mg q2w | Placebo (for Dupilumab 300 mg) q2w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 317 | 631 | 321 | 633
liter
  Baseline | 1.76 (0.61) | 1.78 (0.62) | 1.75 (0.57) | 1.78 (0.60)
  Week 12: number analyzed (Participants) | 307 | 611 | 313 | 610
  Week 12 | 1.92 (0.70) | 2.07 (0.76) | 1.93 (0.68) | 2.09 (0.70)
  Change at Week 12: number analyzed (Participants) | 307 | 611 | 313 | 610
  Change at Week 12 | 0.15 (0.36) | 0.28 (0.45) | 0.18 (0.39) | 0.31 (0.43)
Statistical Analysis 1: Comparison: Placebo (for Dupilumab 300 mg) q2w vs Dupilumab 300 mg q2w; Analysis was performed using mixed-effect model with repeated measures (MMRM) model with change from baseline in FEV1 values up to Week 12 as response variable; and treatment, age, sex, baseline height, region, baseline eosinophil strata, baseline ICS dose level, visit, treatment by-visit interaction, baseline FEV1 value and baseline-by-visit interaction as covariates. Here, it is test no. 2 of testing order; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; Least Square (LS) Mean Difference = 0.13, 95% CI 2-sided [0.08 to 0.18] — Dupilumab 300 mg q2w vs Placebo (for Dupilumab 300 mg) q2w
Statistical Analysis 2: Comparison: Placebo (for Dupilumab 200 mg) q2w vs Dupilumab 200 mg q2w; Analysis was performed using MMRM model with change from baseline in FEV1 values up to Week 12 as response variable; and treatment, age, sex, baseline height, region, baseline eosinophil strata, baseline ICS dose level, visit, treatment by-visit interaction, baseline FEV1 value and baseline-by-visit interaction as covariates. Here, it is test no. 4 of testing order; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = 0.14, 95% CI 2-sided [0.08 to 0.19] — Dupilumab 200 mg q2w vs Placebo (for Dupilumab 200 mg) q2w

3. Secondary Outcome: Percent Change From Baseline in Pre-Bronchodilator FEV1 at Week 12: ITT Population
Description: FEV1 was the volume of air exhaled in the first second of a forced expiration as measured by spirometer.
Time Frame: Baseline, Week 12
Population: Analysis was performed on ITT population. 'Overall number of participants analyzed'=participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo (for Dupilumab 200 mg) q2w | Dupilumab 200 mg q2w | Placebo (for Dupilumab 300 mg) q2w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 307 | 611 | 313 | 610
percent change | 10.16 (23.88) | 18.74 (30.86) | 11.87 (26.40) | 20.89 (34.14)
Statistical Analysis 1: Comparison: Placebo (for Dupilumab 300 mg) q2w vs Dupilumab 300 mg q2w; Analysis performed using MMRM model(n=954 for 300 vs placebo)with percent change from baseline in FEV1 values up to Week 12 as response variable; & treatment, age, sex, baseline height, region, baseline eosinophil strata, baseline ICS dose level, visit, treatment by-visit interaction, baseline FEV1 value & baseline-by-visit interaction as covariates. Hierarchical testing procedure used to control type I error & handle multiple secondary endpoint analyses. Here, it is test no. 5 of testing order; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = 9.41, 95% CI 2-sided [5.74 to 13.07] — Dupilumab 300 mg q2w vs Placebo (for Dupilumab 300 mg) q2w

4. Secondary Outcome: Annualized Rate of Severe Exacerbation Events During The 52-Week Treatment Period: ITT Population With Baseline Eosinophil >=0.15 Giga/L
Description: as for outcome 1
Time Frame: Baseline to Week 52
Population: Analysis was performed ITT population with baseline eosinophil >=0.15 Giga/L.
Measure: Number (95% Confidence Interval); unit: Exacerbation per participant-year
Arm/Group | Placebo (for Dupilumab 200 mg) q2w | Dupilumab 200 mg q2w | Placebo (for Dupilumab 300 mg) q2w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 232 | 437 | 237 | 452
Exacerbation per participant-year | 1.007 [0.814 to 1.245] | 0.445 [0.368 to 0.538] | 1.081 [0.879 to 1.329] | 0.434 [0.359 to 0.525]
Statistical Analysis 1: Comparison: Placebo (for Dupilumab 300 mg) q2w vs Dupilumab 300 mg q2w; Analysis was performed using negative binomial model with total number of events onset from randomization up to Week 52 or last contact date (whichever comes earlier) as response variable; with 4 treatment groups, age, region, baseline eosinophil strata, baseline ICS dose level, number of severe exacerbation events within 1 year prior to study as covariates; and log transformed standardized observation duration as an offset variable. Here, it is test no. 6 of testing order; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.0001, Negative binomial regression model — Threshold for significance at 0.05 level; Relative risk = 0.402, 95% CI 2-sided [0.307 to 0.526] — Dupilumab 300 mg q2w vs Placebo (for Dupilumab 300 mg) q2w

5. Secondary Outcome: Absolute Change From Baseline in Pre-Bronchodilator FEV1 at Week 12: ITT Population With Baseline Eosinophil >=0.15 Giga/L
Description: FEV1 was the volume of air exhaled in the first second of a forced expiration as measured by spirometer.
Time Frame: Baseline, Week 12
Population: Analysis was performed ITT population with baseline eosinophil >=0.15 Giga/L. Here 'Number analyzed' signifies number of participants with available data for specified category.
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | Placebo (for Dupilumab 200 mg) q2w | Dupilumab 200 mg q2w | Placebo (for Dupilumab 300 mg) q2w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 232 | 437 | 237 | 452
liter
  Baseline | 1.77 (0.63) | 1.81 (0.63) | 1.75 (0.55) | 1.79 (0.59)
  Change at Week 12: number analyzed (Participants) | 224 | 425 | 229 | 434
  Change at Week 12 | 0.17 (0.36) | 0.34 (0.46) | 0.21 (0.38) | 0.35 (0.45)
Statistical Analysis 1: Comparison: Placebo (for Dupilumab 300 mg) q2w vs Dupilumab 300 mg q2w; Analysis was performed using MMRM model with change from baseline in FEV1 values up to Week 12 as response variable; and treatment, age, sex, baseline height, region, baseline eosinophil strata, baseline ICS dose level, visit, treatment by-visit interaction, baseline FEV1 value and baseline-by-visit interaction as covariates. Here, it is test no. 7 of testing order; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = 0.15, 95% CI 2-sided [0.09 to 0.21] — Dupilumab 300 mg q2w vs Placebo (for Dupilumab 300 mg) q2w

6. Secondary Outcome: Annualized Rate of Severe Exacerbation Events During The 52-Week Treatment Period: ITT Population With Baseline Eosinophil >=0.3 Giga/L
Description: as for outcome 1
Time Frame: Baseline to Week 52
Population: Analysis was performed on ITT population with baseline eosinophil >=0.3 Giga/L.
Measure: Number (95% Confidence Interval); unit: Exacerbation per participant-year
Arm/Group | Placebo (for Dupilumab 200 mg) q2w | Dupilumab 200 mg q2w | Placebo (for Dupilumab 300 mg) q2w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 148 | 264 | 142 | 277
Exacerbation per participant-year | 1.081 [0.846 to 1.382] | 0.370 [0.289 to 0.475] | 1.236 [0.972 to 1.571] | 0.403 [0.317 to 0.512]
Statistical Analysis 1: Comparison: Placebo (for Dupilumab 300 mg) q2w vs Dupilumab 300 mg q2w; Analysis was performed using negative binomial model with total number of events onset from randomization up to Week 52 or last contact date (whichever comes earlier) as response variable; with 4 treatment groups, age, region, baseline eosinophil strata, baseline ICS dose level, number of severe exacerbation events within 1 year prior to study as covariates; and log transformed standardized observation duration as an offset variable. Here, it is test no. 8 of testing order; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.0001, Negative binomial regression model — Threshold for significance at 0.05 level; Relative risk = 0.326, 95% CI 2-sided [0.234 to 0.454] — Dupilumab 300 mg q2w vs Placebo (for Dupilumab 300 mg) q2w

7. Secondary Outcome: Absolute Change From Baseline in Pre-Bronchodilator FEV1 at Week 12: ITT Population With Baseline Eosinophil >=0.3 Giga/L
Description: FEV1 was the volume of air exhaled in the first second of a forced expiration as measured by spirometer.
Time Frame: Baseline, Week 12
Population: Analysis was performed ITT population with baseline eosinophil >=0.3 Giga/L. Here 'Number analyzed' signifies number of participants with available data for specified category.
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | Placebo (for Dupilumab 200 mg) q2w | Dupilumab 200 mg q2w | Placebo (for Dupilumab 300 mg) q2w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 148 | 264 | 142 | 277
liter
  Baseline | 1.78 (0.66) | 1.81 (0.64) | 1.73 (0.54) | 1.75 (0.59)
  Change at Week 12: number analyzed (Participants) | 144 | 256 | 139 | 266
  Change at Week 12 | 0.19 (0.39) | 0.39 (0.45) | 0.20 (0.40) | 0.43 (0.43)
Statistical Analysis 1: Comparison: Placebo (for Dupilumab 300 mg) q2w vs Dupilumab 300 mg q2w; Analysis was performed using MMRM model with change from baseline in FEV1 values up to Week 12 as response variable; and treatment, age, sex, baseline height, region, baseline eosinophil strata, baseline ICS dose level, visit, treatment by-visit interaction, baseline FEV1 value and baseline-by-visit interaction as covariates. Here, it is test no. 9 of testing order; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = 0.24, 95% CI 2-sided [0.16 to 0.32] — Dupilumab 300 mg q2w vs Placebo (for Dupilumab 300 mg) q2w

8. Secondary Outcome: Annualized Rate of Severe Exacerbation Events During The 52-Week Treatment Period: ITT Population With Baseline Eosinophil <0.3 Giga/L
Description: as for outcome 1
Time Frame: Baseline to Week 52
Population: Analysis was performed on ITT population with baseline eosinophil <0.3 Giga/L.
Measure: Number (95% Confidence Interval); unit: Exacerbation per participant-year
Arm/Group | Placebo (for Dupilumab 200 mg) q2w | Dupilumab 200 mg q2w | Placebo (for Dupilumab 300 mg) q2w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 169 | 366 | 178 | 356
Exacerbation per participant-year | 0.675 [0.515 to 0.884] | 0.512 [0.418 to 0.628] | 0.732 [0.562 to 0.954] | 0.610 [0.502 to 0.742]
Statistical Analysis 1: Comparison: Placebo (for Dupilumab 300 mg) q2w vs Dupilumab 300 mg q2w; Analysis was performed using negative binomial model with total number of events onset from randomization up to Week 52 or last contact date (whichever comes earlier) as response variable; with 4 treatment groups, age, region, baseline eosinophil strata, baseline ICS dose level, number of severe exacerbation events within 1 year prior to study as covariates; and log transformed standardized observation duration as an offset variable. Here, it is test no. 10 of testing order; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p = 0.2599, Negative binomial regression model — Threshold for significance at 0.05 level; Relative risk = 0.834, 95% CI 2-sided [0.608 to 1.144] — Dupilumab 300 mg q2w vs Placebo (for Dupilumab 300 mg) q2w

9. Secondary Outcome: Annualized Rate of Severe Exacerbation Events During The 52-Week Treatment Period: ITT Population With High Dose ICS at Baseline
Description: as for outcome 1
Time Frame: Baseline to Week 52
Population: Analysis was performed on ITT population with high dose ICS at baseline.
Measure: Number (95% Confidence Interval); unit: Exacerbation per participant-year
Arm/Group | Placebo (for Dupilumab 200 mg) q2w | Dupilumab 200 mg q2w | Placebo (for Dupilumab 300 mg) q2w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 172 | 317 | 167 | 323
Exacerbation per participant-year | 1.040 [0.824 to 1.314] | 0.560 [0.455 to 0.690] | 1.038 [0.818 to 1.317] | 0.639 [0.523 to 0.780]

10. Secondary Outcome: Absolute Change From Baseline in Pre-Bronchodilator FEV1 at Week 12: ITT Population With High Dose ICS at Baseline
Description: FEV1 was the volume of air exhaled in the first second of a forced expiration as measured by spirometer.
Time Frame: Baseline, Week 12
Population: Analysis was performed on ITT population with high dose ICS at baseline. 'Overall number of participants analysed'=participants evaluable for this outcome measure at specified timepoint.
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | Placebo (for Dupilumab 200 mg) q2w | Dupilumab 200 mg q2w | Placebo (for Dupilumab 300 mg) q2w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 167 | 310 | 162 | 309
liter | 0.14 (0.34) | 0.27 (0.42) | 0.20 (0.40) | 0.32 (0.43)

11. Secondary Outcome: Change From Baseline in Asthma Quality of Life Questionnaire With Standardized Activities (AQLQ [S]) Self-Administered Global Score at Week 24: ITT Population
Description: The AQLQ is a disease-specific, self-administered quality of life questionnaire designed to measure functional impairments that are most important to participants with asthma. The AQLQ comprises of 32 items in 4 domains: symptoms (12 items), activity limitation (11 items), emotional function (5 items), environmental stimuli (4 items). Each item is scored on a 7-point likert scale (1=maximal impairment, 7=no impairment). The 32 items of the questionnaire are averaged to produce one overall quality of life score ranging from 1 (severely impaired) to 7 (not impaired at all). Higher scores indicate better quality of life.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo (for Dupilumab 200 mg) q2w | Dupilumab 200 mg q2w | Placebo (for Dupilumab 300 mg) q2w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 317 | 631 | 321 | 633
scores on a scale
  Baseline: number analyzed (Participants) | 299 | 591 | 314 | 603
  Baseline | 4.26 (1.02) | 4.31 (1.08) | 4.30 (1.03) | 4.28 (1.05)
  Week 24: number analyzed (Participants) | 298 | 592 | 302 | 596
  Week 24 | 5.23 (1.07) | 5.46 (1.12) | 5.30 (1.15) | 5.47 (1.09)
  Change at Week 24: number analyzed (Participants) | 281 | 560 | 295 | 569
  Change at Week 24 | 0.95 (1.03) | 1.13 (1.14) | 1.02 (1.10) | 1.17 (1.11)

12. Secondary Outcome: Change From Baseline in AQLQ (S) Self- Administered Global Score at Week 24: ITT Population With Baseline Eosinophil >=0.3 Giga/L
Description: as for outcome 11
Time Frame: Baseline, Week 24
Population: Analysis was performed on ITT population with baseline eosinophil >=0.3 Giga/L. Here 'Number analyzed' signifies number of participants with available data for specified category.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo (for Dupilumab 200 mg) q2w | Dupilumab 200 mg q2w | Placebo (for Dupilumab 300 mg) q2w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 148 | 264 | 142 | 277
scores on a scale
  Baseline: number analyzed (Participants) | 136 | 254 | 138 | 263
  Baseline | 4.24 (0.98) | 4.24 (1.11) | 4.21 (0.97) | 4.36 (1.05)
  Change at Week 24: number analyzed (Participants) | 129 | 241 | 130 | 244
  Change at Week 24 | 0.97 (1.01) | 1.39 (1.15) | 1.02 (1.25) | 1.30 (1.15)

13. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire 5-item Version (ACQ-5) Score at Week 24: ITT Population
Description: The ACQ-5 has 5 questions, reflecting the top-scoring five asthma symptoms: woken at night by symptoms, wake in the mornings with symptoms, limitation of daily activities, shortness of breath and wheeze. Participants were asked to recall how their asthma had been during the previous week and to respond to each of the five symptom questions on a 7-point scale ranged from 0 (no impairment) to 6 (maximum impairment). ACQ-5 total score was mean of the scores of all 5 questions and, therefore, ranged from 0 (totally controlled) to 6 (severely uncontrolled). Higher score indicated lower asthma control.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo (for Dupilumab 200 mg) q2w | Dupilumab 200 mg q2w | Placebo (for Dupilumab 300 mg) q2w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 317 | 631 | 321 | 633
scores on a scale
  Baseline | 2.71 (0.73) | 2.76 (0.80) | 2.77 (0.77) | 2.77 (0.76)
  Week 24: number analyzed (Participants) | 296 | 590 | 297 | 585
  Week 24 | 1.67 (1.06) | 1.33 (1.05) | 1.58 (1.08) | 1.37 (1.10)
  Change at Week 24: number analyzed (Participants) | 296 | 590 | 297 | 585
  Change at Week 24 | -1.06 (1.01) | -1.43 (1.05) | -1.19 (1.10) | -1.38 (1.10)

14. Secondary Outcome: Annualized Rate of Severe Exacerbation Events Resulting in Hospitalization or Emergency Room Visit During The 52-Week Treatment Period: ITT Population
Description: A severe exacerbation was defined as a deterioration of asthma requiring: use of systemic corticosteroids for >=3 days; or hospitalization or emergency room visit because of asthma, requiring systemic corticosteroids. Annualized event rate was the total number of exacerbations (resulted hospitalization or emergency room visit) that occurred during the treatment period divided by the total number of participant-years treated.
Time Frame: Baseline to Week 52
Population: Analysis was performed on ITT population.
Measure: Number (95% Confidence Interval); unit: Exacerbation per participant-year
Arm/Group | Placebo (for Dupilumab 200 mg) q2w | Dupilumab 200 mg q2w | Placebo (for Dupilumab 300 mg) q2w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 317 | 631 | 321 | 633
Exacerbation per participant-year | 0.081 [0.049 to 0.135] | 0.043 [0.027 to 0.068] | 0.034 [0.017 to 0.066] | 0.025 [0.014 to 0.043]

15. Secondary Outcome: Absolute Change From Baseline in Pre-Bronchodilator FEV1 at Week 12: ITT Population With Baseline Eosinophil <0.3 Giga/L
Description: FEV1 was the volume of air exhaled in the first second of a forced expiration as measured by spirometer.
Time Frame: Baseline, Week 12
Population: Analysis was performed ITT population with baseline eosinophil <0.3 Giga/L. 'Overall number of participants analysed'=participants evaluable for this outcome measure at specified timepoint.
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | Placebo (for Dupilumab 200 mg) q2w | Dupilumab 200 mg q2w | Placebo (for Dupilumab 300 mg) q2w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 163 | 354 | 173 | 344
liter | 0.12 (0.32) | 0.21 (0.43) | 0.17 (0.39) | 0.21 (0.41)

16. Secondary Outcome: Percent Change From Baseline in Pre-Bronchodilator FEV1 at Week 12: ITT Population With Baseline Eosinophil >=0.3 Giga/L
Description: FEV1 was the volume of air exhaled in the first second of a forced expiration as measured by spirometer.
Time Frame: Baseline, Week 12
Population: Analysis was performed on ITT population with baseline eosinophil >=0.3 Giga/L. 'Overall number of participants analyzed'=participants evaluable for this outcome measure at specified timepoint.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo (for Dupilumab 200 mg) q2w | Dupilumab 200 mg q2w | Placebo (for Dupilumab 300 mg) q2w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 144 | 256 | 139 | 266
percent change | 13.40 (27.01) | 26.41 (33.69) | 13.05 (25.27) | 30.58 (38.22)

17. Secondary Outcome: Percent Change From Baseline in Pre-Bronchodilator FEV1 at Week 12: ITT Population With High Dose ICS at Baseline
Description: FEV1 was the volume of air exhaled in the first second of a forced expiration as measured by spirometer.
Time Frame: Baseline, Week 12
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo (for Dupilumab 200 mg) q2w | Dupilumab 200 mg q2w | Placebo (for Dupilumab 300 mg) q2w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 167 | 310 | 162 | 309
percent change | 8.47 (20.94) | 17.99 (28.43) | 13.22 (26.52) | 23.41 (37.26)

18. Secondary Outcome: Percent Change From Baseline in Pre-Bronchodilator FEV1 at Week 12: ITT Population With Baseline Eosinophil >=0.15 Giga/L
Description: FEV1 was the volume of air exhaled in the first second of a forced expiration as measured by spirometer.
Time Frame: Baseline, Week 12
Population: Analysis was performed on ITT population with baseline eosinophil >=0.15 Giga/L. 'Overall number of participants analyzed'=participants evaluable for this outcome measure at specified timepoint.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo (for Dupilumab 200 mg) q2w | Dupilumab 200 mg q2w | Placebo (for Dupilumab 300 mg) q2w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 224 | 425 | 229 | 434
percent change | 11.43 (24.71) | 22.04 (31.96) | 13.49 (25.18) | 24.04 (35.71)

19. Secondary Outcome: Absolute Change From Baseline in Pre-Bronchodilator FEV1 at Weeks 2, 4, 8, 24, 36, and 52: ITT Population
Description: FEV1 was the volume of air exhaled in the first second of a forced expiration as measured by spirometer.
Time Frame: Baseline, Weeks 2, 4, 8, 24, 36, and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | Placebo (for Dupilumab 200 mg) q2w | Dupilumab 200 mg q2w | Placebo (for Dupilumab 300 mg) q2w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 317 | 631 | 321 | 633
liter
  Change at Week 2: number analyzed (Participants) | 315 | 610 | 313 | 625
  Change at Week 2 | 0.08 (0.35) | 0.22 (0.38) | 0.10 (0.34) | 0.25 (0.40)
  Change at Week 4: number analyzed (Participants) | 307 | 613 | 311 | 614
  Change at Week 4 | 0.13 (0.35) | 0.24 (0.40) | 0.13 (0.34) | 0.27 (0.41)
  Change at Week 8: number analyzed (Participants) | 305 | 604 | 311 | 609
  Change at Week 8 | 0.15 (0.38) | 0.28 (0.42) | 0.19 (0.40) | 0.29 (0.43)
  Change at Week 24: number analyzed (Participants) | 300 | 599 | 296 | 596
  Change at Week 24 | 0.13 (0.40) | 0.31 (0.45) | 0.19 (0.44) | 0.30 (0.44)
  Change at Week 36: number analyzed (Participants) | 289 | 590 | 301 | 584
  Change at Week 36 | 0.14 (0.41) | 0.31 (0.48) | 0.21 (0.42) | 0.32 (0.45)
  Change at Week 52: number analyzed (Participants) | 240 | 477 | 250 | 488
  Change at Week 52 | 0.12 (0.38) | 0.31 (0.50) | 0.20 (0.42) | 0.32 (0.44)

20. Secondary Outcome: Percent Change From Baseline in Pre-Bronchodilator FEV1 at Weeks 2, 4, 8, 24, 36, and 52: ITT Population
Description: FEV1 was the volume of air exhaled in the first second of a forced expiration as measured by spirometer.
Time Frame: Baseline, Weeks 2, 4, 8, 24, 36, and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo (for Dupilumab 200 mg) q2w | Dupilumab 200 mg q2w | Placebo (for Dupilumab 300 mg) q2w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 317 | 631 | 321 | 633
percent change
  Change at Week 2: number analyzed (Participants) | 315 | 610 | 313 | 625
  Change at Week 2 | 5.78 (23.36) | 14.32 (26.55) | 6.60 (21.84) | 17.38 (30.82)
  Change at Week 4: number analyzed (Participants) | 307 | 613 | 311 | 614
  Change at Week 4 | 9.61 (25.54) | 16.11 (28.12) | 8.67 (23.55) | 18.77 (32.73)
  Change at Week 8: number analyzed (Participants) | 305 | 604 | 311 | 609
  Change at Week 8 | 10.27 (25.60) | 18.81 (29.80) | 12.24 (25.78) | 19.85 (33.63)
  Change at Week 24: number analyzed (Participants) | 300 | 599 | 296 | 596
  Change at Week 24 | 9.42 (26.76) | 19.76 (30.64) | 12.86 (28.14) | 20.75 (35.35)
  Change at Week 36: number analyzed (Participants) | 289 | 590 | 301 | 584
  Change at Week 36 | 10.57 (26.41) | 19.92 (32.26) | 13.45 (27.69) | 22.08 (35.93)
  Change at Week 52: number analyzed (Participants) | 240 | 477 | 250 | 488
  Change at Week 52 | 8.37 (23.59) | 19.96 (33.35) | 12.89 (27.70) | 21.57 (34.08)

21. Secondary Outcome: Change From Baseline in Percent Predicted FEV1 at Weeks 2, 4, 8, 12, 24, 36, and 52: ITT Population
Description: FEV1 was the volume of air exhaled in the first second of a forced expiration as measured by spirometer.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 24, 36, and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent predicted of FEV1
Arm/Group | Placebo (for Dupilumab 200 mg) q2w | Dupilumab 200 mg q2w | Placebo (for Dupilumab 300 mg) q2w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 317 | 631 | 321 | 633
percent predicted of FEV1
  Change at Week 2: number analyzed (Participants) | 315 | 610 | 313 | 625
  Change at Week 2 | 2.58 (11.36) | 7.10 (12.28) | 3.32 (10.98) | 8.44 (13.20)
  Change at Week 4: number analyzed (Participants) | 307 | 613 | 311 | 614
  Change at Week 4 | 4.55 (11.69) | 7.92 (12.81) | 4.13 (11.41) | 9.20 (14.10)
  Change at Week 8: number analyzed (Participants) | 305 | 604 | 311 | 609
  Change at Week 8 | 4.93 (12.30) | 9.27 (13.13) | 6.08 (12.55) | 9.70 (14.15)
  Change at Week 12: number analyzed (Participants) | 307 | 611 | 313 | 610
  Change at Week 12 | 5.02 (12.10) | 9.22 (13.87) | 5.90 (13.02) | 10.28 (14.44)
  Change at Week 24: number analyzed (Participants) | 300 | 599 | 296 | 596
  Change at Week 24 | 4.38 (12.85) | 9.98 (13.94) | 6.41 (14.02) | 10.14 (14.75)
  Change at Week 36: number analyzed (Participants) | 289 | 590 | 301 | 584
  Change at Week 36 | 5.09 (12.99) | 10.12 (14.61) | 6.82 (13.54) | 10.94 (15.06)
  Change at Week 52: number analyzed (Participants) | 240 | 477 | 250 | 488
  Change at Week 52 | 4.25 (12.06) | 10.08 (14.79) | 6.68 (13.56) | 11.02 (14.59)

22. Secondary Outcome: Change From Baseline in Morning (AM)/Evening (PM) Peak Expiratory Flow (PEF) at Weeks 2, 4, 8, 12, 24, 36, and 52: ITT Population
Description: The PEF is a participant's maximum speed of expiration, as measured with a peak flow meter. Peak flow testing for PEF was performed at home (morning and evening) while sitting or standing prior to using any medication (if needed) for asthma.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 24, 36, and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: liters/min
Arm/Group | Placebo (for Dupilumab 200 mg) q2w | Dupilumab 200 mg q2w | Placebo (for Dupilumab 300 mg) q2w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 317 | 631 | 321 | 633
liters/min
  AM: Change at Week 2: number analyzed (Participants) | 314 | 620 | 320 | 630
  AM: Change at Week 2 | 4.19 (31.30) | 15.21 (39.45) | 3.45 (28.95) | 14.46 (36.29)
  AM: Change at Week 4: number analyzed (Participants) | 313 | 619 | 319 | 625
  AM: Change at Week 4 | 6.23 (42.42) | 21.81 (53.85) | 5.55 (43.69) | 19.67 (46.47)
  AM: Change at Week 8: number analyzed (Participants) | 308 | 614 | 318 | 613
  AM: Change at Week 8 | 7.42 (49.30) | 25.70 (58.52) | 12.22 (50.50) | 23.18 (52.65)
  AM: Change at Week 12: number analyzed (Participants) | 305 | 608 | 314 | 608
  AM: Change at Week 12 | 9.85 (50.40) | 27.81 (65.30) | 14.23 (56.18) | 25.88 (57.09)
  AM: Change at Week 24: number analyzed (Participants) | 299 | 590 | 305 | 588
  AM: Change at Week 24 | 5.55 (53.27) | 28.71 (69.64) | 15.43 (60.83) | 23.74 (63.71)
  AM: Change at Week 36: number analyzed (Participants) | 289 | 576 | 297 | 564
  AM: Change at Week 36 | 3.24 (61.68) | 31.19 (71.59) | 12.57 (61.88) | 23.93 (65.04)
  AM: Change at Week 52: number analyzed (Participants) | 270 | 544 | 282 | 529
  AM: Change at Week 52 | 2.85 (64.60) | 29.86 (75.44) | 10.99 (64.68) | 26.67 (71.63)
  PM: Change at Week 2: number analyzed (Participants) | 313 | 617 | 319 | 629
  PM: Change at Week 2 | 3.33 (36.81) | 13.80 (40.59) | 3.87 (33.98) | 11.35 (36.10)
  PM: Change at Week 4: number analyzed (Participants) | 312 | 617 | 319 | 623
  PM: Change at Week 4 | 5.01 (45.09) | 17.94 (55.30) | 2.73 (46.83) | 14.90 (47.42)
  PM: Change at Week 8: number analyzed (Participants) | 308 | 613 | 315 | 610
  PM: Change at Week 8 | 2.82 (50.10) | 21.06 (61.80) | 7.68 (56.73) | 17.26 (53.37)
  PM: Change at Week 12: number analyzed (Participants) | 306 | 606 | 311 | 605
  PM: Change at Week 12 | 3.24 (53.42) | 19.75 (68.14) | 8.52 (56.74) | 18.70 (55.60)
  PM: Change at Week 24: number analyzed (Participants) | 299 | 583 | 300 | 585
  PM: Change at Week 24 | -4.89 (55.07) | 19.95 (71.50) | 7.56 (63.25) | 15.82 (61.91)
  PM: Change at Week 36: number analyzed (Participants) | 286 | 570 | 291 | 557
  PM: Change at Week 36 | -6.75 (62.44) | 21.79 (75.00) | 2.64 (65.21) | 14.35 (64.66)
  PM: Change at Week 52: number analyzed (Participants) | 269 | 526 | 268 | 523
  PM: Change at Week 52 | -6.43 (62.82) | 18.77 (77.37) | 2.83 (67.01) | 15.58 (72.51)

23. Secondary Outcome: Change From Baseline in Forced Vital Capacity (FVC) at Weeks 2, 4, 8, 12, 24, 36, and 52: ITT Population
Description: FVC is a standard pulmonary function test used to quantify respiratory muscle weakness. FVC is the volume of air that can forcibly be blown out after full inspiration in the upright position, measured in liters.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 24, 36, and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | Placebo (for Dupilumab 200 mg) q2w | Dupilumab 200 mg q2w | Placebo (for Dupilumab 300 mg) q2w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 317 | 631 | 321 | 633
liter
  Change at Week 2: number analyzed (Participants) | 315 | 610 | 313 | 625
  Change at Week 2 | 0.08 (0.42) | 0.23 (0.44) | 0.10 (0.37) | 0.25 (0.46)
  Change at Week 4: number analyzed (Participants) | 307 | 613 | 311 | 614
  Change at Week 4 | 0.12 (0.39) | 0.26 (0.45) | 0.12 (0.38) | 0.27 (0.47)
  Change at Week 8: number analyzed (Participants) | 305 | 604 | 311 | 609
  Change at Week 8 | 0.13 (0.41) | 0.28 (0.45) | 0.18 (0.42) | 0.29 (0.50)
  Change at Week 12: number analyzed (Participants) | 307 | 611 | 313 | 610
  Change at Week 12 | 0.13 (0.41) | 0.29 (0.49) | 0.18 (0.44) | 0.29 (0.51)
  Change at Week 24: number analyzed (Participants) | 300 | 599 | 296 | 596
  Change at Week 24 | 0.11 (0.45) | 0.29 (0.48) | 0.18 (0.46) | 0.29 (0.51)
  Change at Week 36: number analyzed (Participants) | 289 | 590 | 301 | 584
  Change at Week 36 | 0.11 (0.45) | 0.30 (0.52) | 0.19 (0.47) | 0.31 (0.52)
  Change at Week 52: number analyzed (Participants) | 240 | 477 | 250 | 488
  Change at Week 52 | 0.08 (0.45) | 0.29 (0.53) | 0.18 (0.45) | 0.31 (0.50)

24. Secondary Outcome: Change From Baseline in Forced Expiratory Flow (FEF) 25-75% at Weeks 2, 4, 8, 12, 24, 36, and 52: ITT Population
Description: FEF is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation. FEF25-75% is defined as the mean forced expiratory flow between the 25% and 75% of the FVC.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 24, 36, and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: liters/sec
Arm/Group | Placebo (for Dupilumab 200 mg) q2w | Dupilumab 200 mg q2w | Placebo (for Dupilumab 300 mg) q2w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 317 | 631 | 321 | 633
liters/sec
  Change at Week 2: number analyzed (Participants) | 315 | 610 | 313 | 625
  Change at Week 2 | 0.09 (0.40) | 0.22 (0.47) | 0.11 (0.44) | 0.27 (0.48)
  Change at Week 4: number analyzed (Participants) | 307 | 613 | 311 | 614
  Change at Week 4 | 0.16 (0.45) | 0.24 (0.48) | 0.15 (0.44) | 0.29 (0.48)
  Change at Week 8: number analyzed (Participants) | 305 | 604 | 311 | 609
  Change at Week 8 | 0.18 (0.45) | 0.29 (0.52) | 0.20 (0.49) | 0.32 (0.51)
  Change at Week 12: number analyzed (Participants) | 307 | 611 | 313 | 610
  Change at Week 12 | 0.18 (0.46) | 0.30 (0.53) | 0.19 (0.50) | 0.35 (0.53)
  Change at Week 24: number analyzed (Participants) | 300 | 599 | 296 | 596
  Change at Week 24 | 0.17 (0.47) | 0.34 (0.57) | 0.22 (0.56) | 0.35 (0.54)
  Change at Week 36: number analyzed (Participants) | 289 | 590 | 301 | 584
  Change at Week 36 | 0.18 (0.49) | 0.35 (0.59) | 0.22 (0.49) | 0.36 (0.56)
  Change at Week 52: number analyzed (Participants) | 240 | 477 | 250 | 488
  Change at Week 52 | 0.16 (0.50) | 0.36 (0.63) | 0.24 (0.55) | 0.36 (0.55)

25. Secondary Outcome: Change From Baseline in Post-Bronchodilator FEV1 at Weeks 2, 4, 8, 12, 24, 36, and 52: ITT Population
Description: FEV1 was the volume of air exhaled in the first second of a forced expiration as measured by spirometer.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 24, 36, and 52
Population: Analysis was performed ITT population. Here 'Number analyzed' signifies number of participants with available data for specified category.
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | Placebo (for Dupilumab 200 mg) q2w | Dupilumab 200 mg q2w | Placebo (for Dupilumab 300 mg) q2w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 317 | 631 | 321 | 633
liter
  Change at Week 2: number analyzed (Participants) | 310 | 609 | 311 | 617
  Change at Week 2 | -0.07 (0.31) | 0.10 (0.37) | -0.04 (0.33) | 0.09 (0.34)
  Change at Week 4: number analyzed (Participants) | 308 | 614 | 311 | 615
  Change at Week 4 | -0.02 (0.31) | 0.10 (0.39) | -0.04 (0.36) | 0.10 (0.36)
  Change at Week 8: number analyzed (Participants) | 305 | 607 | 305 | 604
  Change at Week 8 | -0.02 (0.31) | 0.12 (0.40) | 0.03 (0.35) | 0.11 (0.37)
  Change at Week 12: number analyzed (Participants) | 305 | 610 | 313 | 612
  Change at Week 12 | -0.02 (0.33) | 0.12 (0.40) | 0.01 (0.35) | 0.11 (0.38)
  Change at Week 24: number analyzed (Participants) | 302 | 599 | 302 | 601
  Change at Week 24 | -0.05 (0.36) | 0.13 (0.43) | -0.01 (0.40) | 0.10 (0.39)
  Change at Week 36: number analyzed (Participants) | 290 | 586 | 302 | 589
  Change at Week 36 | -0.03 (0.34) | 0.12 (0.44) | 0.01 (0.38) | 0.11 (0.39)
  Change at Week 52: number analyzed (Participants) | 239 | 499 | 255 | 494
  Change at Week 52 | -0.08 (0.38) | 0.12 (0.44) | -0.02 (0.39) | 0.11 (0.40)

26. Secondary Outcome: Annualized Rate of Loss of Asthma Control (LOAC) Event During The 52-Week Treatment Period: ITT Population
Description: LOAC was defined as any of the following: >=6 additional reliever puffs of salbutamol/albuterol or levosalbutamol/levalbuterol in a 24-hour period (compared to baseline) on 2 consecutive days; increase in ICS >=4 times the dose at randomization; use of systemic corticosteroids for >=3 days; hospitalization or emergency room visit because of asthma, requiring systemic corticosteroids. Annualized event rate was the total number of LOAC that occurred during the treatment period divided by the total number of participant-years treated.
Time Frame: Baseline to Week 52
Population: Analysis was performed on ITT population.
Measure: Number (95% Confidence Interval); unit: LOAC per participant-year
Arm/Group | Placebo (for Dupilumab 200 mg) q2w | Dupilumab 200 mg q2w | Placebo (for Dupilumab 300 mg) q2w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 317 | 631 | 321 | 633
LOAC per participant-year | 2.972 [2.573 to 3.432] | 1.853 [1.654 to 2.076] | 2.965 [2.572 to 3.420] | 1.740 [1.554 to 1.947]

27. Secondary Outcome: Time to First Severe Exacerbation Event: Kaplan-Meier Estimates During The 52-Week Treatment Period: ITT Population
Description: The time to first severe exacerbation was defined as follows: date of the first event - randomization date +1. For participants who had no event on or before Visit 18 (Week 52) or last contact date, the time was censored at the date of Visit 18 or the last contact date, whichever was earlier. The median time to first severe exacerbation was not estimated; therefore, the probability of severe exacerbation at Weeks 12, 24, 36, and 52, are presented as the descriptive statistics.
Time Frame: Baseline up to Week 52
Population: Analysis was performed on ITT population.
Measure: Number (95% Confidence Interval); unit: probability of severe exacerbation
Arm/Group | Placebo (for Dupilumab 200 mg) q2w | Dupilumab 200 mg q2w | Placebo (for Dupilumab 300 mg) q2w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 317 | 631 | 321 | 633
probability of severe exacerbation
  Probability at Week 12 | 0.165 [0.127 to 0.209] | 0.094 [0.073 to 0.119] | 0.193 [0.152 to 0.238] | 0.137 [0.112 to 0.166]
  Probability at Week 24 | 0.275 [0.227 to 0.326] | 0.177 [0.148 to 0.208] | 0.297 [0.247 to 0.347] | 0.211 [0.180 to 0.243]
  Probability at Week 36 | 0.364 [0.311 to 0.418] | 0.235 [0.203 to 0.270] | 0.376 [0.322 to 0.428] | 0.268 [0.234 to 0.303]
  Probability at Week 52 | 0.434 [0.378 to 0.489] | 0.295 [0.259 to 0.331] | 0.437 [0.382 to 0.491] | 0.325 [0.288 to 0.362]

28. Secondary Outcome: Time to First LOAC Event: Kaplan-Meier Estimates During The 52-Week Treatment Period: ITT Population
Description: The time to first LOAC event was defined as follows: date of the first event - first dose date +1. For participants who had no event on or before last dose date + 14 days or last contact date, the time was censored at the last dose date + 14 days or the last contact date, whichever was earlier.
Time Frame: Baseline up to Week 52
Population: Analysis was performed on ITT population.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo (for Dupilumab 200 mg) q2w | Dupilumab 200 mg q2w | Placebo (for Dupilumab 300 mg) q2w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 317 | 631 | 321 | 633
days | 110.0 [84.00 to 144.00] | 230.0 [187.00 to 276.00] | 102.0 [74.00 to 130.00] | 264.0 [207.00 to 319.00]

29. Secondary Outcome: Change From Baseline in ACQ-5 Score at Weeks 2, 4, 8, 12, 36, and 52: ITT Population
Description: as for outcome 13
Time Frame: Baseline, Weeks 2, 4, 8, 12, 36, and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo (for Dupilumab 200 mg) q2w | Dupilumab 200 mg q2w | Placebo (for Dupilumab 300 mg) q2w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 317 | 631 | 321 | 633
scores on a scale
  Change at Week 2: number analyzed (Participants) | 304 | 599 | 305 | 615
  Change at Week 2 | -0.52 (0.85) | -0.88 (0.91) | -0.58 (0.97) | -0.89 (0.94)
  Change at Week 4: number analyzed (Participants) | 297 | 599 | 305 | 605
  Change at Week 4 | -0.76 (0.90) | -1.07 (0.98) | -0.77 (1.01) | -1.06 (1.01)
  Change at Week 8: number analyzed (Participants) | 301 | 595 | 310 | 593
  Change at Week 8 | -0.94 (0.96) | -1.26 (1.03) | -1.05 (1.04) | -1.24 (1.06)
  Change at Week 12: number analyzed (Participants) | 303 | 605 | 312 | 603
  Change at Week 12 | -0.98 (1.00) | -1.33 (1.03) | -1.09 (1.09) | -1.35 (1.06)
  Change at Week 36: number analyzed (Participants) | 285 | 583 | 299 | 572
  Change at Week 36 | -1.21 (1.01) | -1.50 (1.14) | -1.22 (1.09) | -1.52 (1.09)
  Change at Week 52: number analyzed (Participants) | 236 | 470 | 245 | 477
  Change at Week 52 | -1.07 (1.08) | -1.50 (1.05) | -1.25 (1.05) | -1.50 (1.08)

30. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire 7-item Version (ACQ-7) Score at Weeks 2, 4, 8, 12, 24, 36, and 52: ITT Population
Description: The ACQ-7 has 7 questions, the first 5 questions assess the most common asthma symptoms: woken at night by symptoms, wake in the mornings with symptoms, limitation of daily activities, shortness of breath and wheeze plus short-acting bronchodilator use, and FEV1 (pre-bronchodilator % predicted). Participants were asked to recall how their asthma had been during the previous week and to respond to each of the five symptom questions on a 7-point scale ranged from 0 (no impairment) to 6 (maximum impairment). Clinic staff scored the FEV1% predicted on a 7-point scale. The questions were equally weighted and the ACQ-7 total score was mean of the scores of all 7 questions and, therefore, ranged from 0 (totally controlled) to 6 (severely uncontrolled). Higher score indicated lower asthma control.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 24, 36, and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo (for Dupilumab 200 mg) q2w | Dupilumab 200 mg q2w | Placebo (for Dupilumab 300 mg) q2w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 317 | 631 | 321 | 633
scores on a scale
  Change at Week 2: number analyzed (Participants) | 304 | 599 | 305 | 615
  Change at Week 2 | -0.46 (0.70) | -0.79 (0.77) | -0.50 (0.80) | -0.82 (0.81)
  Change at Week 4: number analyzed (Participants) | 297 | 599 | 305 | 605
  Change at Week 4 | -0.65 (0.76) | -0.94 (0.85) | -0.65 (0.85) | -0.97 (0.87)
  Change at Week 8: number analyzed (Participants) | 301 | 595 | 310 | 593
  Change at Week 8 | -0.81 (0.80) | -1.11 (0.90) | -0.90 (0.89) | -1.12 (0.92)
  Change at Week 12: number analyzed (Participants) | 303 | 605 | 312 | 603
  Change at Week 12 | -0.85 (0.83) | -1.17 (0.90) | -0.92 (0.93) | -1.20 (0.92)
  Change at Week 24: number analyzed (Participants) | 296 | 590 | 297 | 585
  Change at Week 24 | -0.89 (0.91) | -1.25 (0.92) | -1.01 (0.96) | -1.22 (0.96)
  Change at Week 36: number analyzed (Participants) | 285 | 583 | 299 | 572
  Change at Week 36 | -1.04 (0.84) | -1.32 (1.01) | -1.05 (0.94) | -1.35 (0.95)
  Change at Week 52: number analyzed (Participants) | 236 | 470 | 245 | 477
  Change at Week 52 | -0.91 (0.92) | -1.32 (0.91) | -1.07 (0.91) | -1.34 (0.93)

31. Secondary Outcome: Change From Baseline in Morning Asthma Symptom Score at Weeks 2, 4, 8, 12, 24, 36, and 52: ITT Population
Description: Morning asthma symptom score was determined using AM (ante meridiem) symptom scoring system which evaluated participant's overall asthma symptoms experienced during the night. It ranged from 0 to 4 as: 0= No asthma symptoms, slept through the night, 1= Slept well, but some complaints in the morning, no night time awakenings, 2= Woke up once because of asthma (including early awakening), 3= Woke up several times because of asthma (including early awakening), 4= Bad night, awake most of the night because of asthma.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 24, 36, and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo (for Dupilumab 200 mg) q2w | Dupilumab 200 mg q2w | Placebo (for Dupilumab 300 mg) q2w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 317 | 631 | 321 | 633
scores on a scale
  Change at Week 2: number analyzed (Participants) | 314 | 624 | 321 | 631
  Change at Week 2 | -0.07 (0.43) | -0.18 (0.49) | -0.09 (0.49) | -0.15 (0.50)
  Change at Week 4: number analyzed (Participants) | 313 | 623 | 319 | 627
  Change at Week 4 | -0.16 (0.59) | -0.26 (0.59) | -0.16 (0.61) | -0.27 (0.64)
  Change at Week 8: number analyzed (Participants) | 308 | 620 | 318 | 615
  Change at Week 8 | -0.26 (0.64) | -0.40 (0.68) | -0.25 (0.62) | -0.37 (0.70)
  Change at Week 12: number analyzed (Participants) | 306 | 614 | 315 | 609
  Change at Week 12 | -0.30 (0.64) | -0.45 (0.71) | -0.30 (0.69) | -0.44 (0.72)
  Change at Week 24: number analyzed (Participants) | 302 | 602 | 306 | 592
  Change at Week 24 | -0.35 (0.69) | -0.52 (0.76) | -0.36 (0.73) | -0.50 (0.73)
  Change at Week 36: number analyzed (Participants) | 292 | 583 | 299 | 572
  Change at Week 36 | -0.38 (0.69) | -0.54 (0.81) | -0.38 (0.76) | -0.56 (0.77)
  Change at Week 52: number analyzed (Participants) | 275 | 553 | 286 | 540
  Change at Week 52 | -0.41 (0.71) | -0.55 (0.84) | -0.41 (0.78) | -0.60 (0.79)

32. Secondary Outcome: Change From Baseline in Evening Asthma Symptom Score at Weeks 2, 4, 8, 12, 24, 36, and 52: ITT Population
Description: Evening asthma symptom score was determined using PM (post meridiem) symptom scoring system which evaluated participant's overall asthma symptoms experienced during the day. It ranged from 0 to 4 as: 0=very well, no asthma symptoms, 1=one episode of wheezing, cough, or breathlessness, 2=more than one episode of wheezing, cough, or breathlessness without interference of normal activities, 3=wheezing, cough, or breathlessness most of the day, which interfered to some extent with normal activities, 4=asthma very bad, unable to carry out daily activities as usual.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 24, 36, and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo (for Dupilumab 200 mg) q2w | Dupilumab 200 mg q2w | Placebo (for Dupilumab 300 mg) q2w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 317 | 631 | 321 | 633
scores on a scale
  Change at Week 2: number analyzed (Participants) | 313 | 624 | 320 | 631
  Change at Week 2 | -0.05 (0.45) | -0.17 (0.48) | -0.06 (0.45) | -0.16 (0.52)
  Change at Week 4: number analyzed (Participants) | 313 | 623 | 319 | 628
  Change at Week 4 | -0.11 (0.59) | -0.27 (0.61) | -0.14 (0.58) | -0.29 (0.64)
  Change at Week 8: number analyzed (Participants) | 308 | 619 | 318 | 612
  Change at Week 8 | -0.24 (0.64) | -0.41 (0.70) | -0.22 (0.63) | -0.40 (0.70)
  Change at Week 12: number analyzed (Participants) | 307 | 612 | 314 | 606
  Change at Week 12 | -0.26 (0.66) | -0.45 (0.72) | -0.30 (0.68) | -0.46 (0.73)
  Change at Week 24: number analyzed (Participants) | 301 | 596 | 301 | 590
  Change at Week 24 | -0.33 (0.72) | -0.52 (0.78) | -0.36 (0.72) | -0.52 (0.73)
  Change at Week 36: number analyzed (Participants) | 289 | 576 | 292 | 566
  Change at Week 36 | -0.39 (0.73) | -0.56 (0.81) | -0.39 (0.75) | -0.56 (0.80)
  Change at Week 52: number analyzed (Participants) | 274 | 536 | 270 | 535
  Change at Week 52 | -0.41 (0.74) | -0.57 (0.84) | -0.42 (0.75) | -0.61 (0.78)

33. Secondary Outcome: Change From Baseline in Number of Nocturnal Awakenings Per Night at Weeks 2, 4, 8, 12, 24, 36, and 52: ITT Population
Description: Participants recorded every morning on awakening the number of asthma-related nocturnal awakenings requiring use of rescue medication that occurred during the previous night.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 24, 36, and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: number of nocturnal awakenings/night
Arm/Group | Placebo (for Dupilumab 200 mg) q2w | Dupilumab 200 mg q2w | Placebo (for Dupilumab 300 mg) q2w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 317 | 631 | 321 | 633
number of nocturnal awakenings/night
  Change at Week 2: number analyzed (Participants) | 314 | 624 | 321 | 631
  Change at Week 2 | -0.06 (0.49) | -0.15 (0.55) | -0.04 (0.62) | -0.11 (0.67)
  Change at Week 4: number analyzed (Participants) | 313 | 623 | 319 | 627
  Change at Week 4 | -0.10 (0.61) | -0.19 (0.66) | -0.11 (0.70) | -0.20 (0.67)
  Change at Week 8: number analyzed (Participants) | 308 | 620 | 318 | 615
  Change at Week 8 | -0.18 (0.65) | -0.29 (0.72) | -0.17 (0.62) | -0.24 (0.72)
  Change at Week 12: number analyzed (Participants) | 306 | 614 | 315 | 609
  Change at Week 12 | -0.21 (0.66) | -0.33 (0.75) | -0.18 (0.67) | -0.28 (0.73)
  Change at Week 24: number analyzed (Participants) | 302 | 602 | 306 | 592
  Change at Week 24 | -0.23 (0.78) | -0.36 (0.81) | -0.26 (0.65) | -0.30 (0.73)
  Change at Week 36: number analyzed (Participants) | 292 | 583 | 299 | 572
  Change at Week 36 | -0.25 (0.74) | -0.34 (0.81) | -0.26 (0.71) | -0.36 (0.74)
  Change at Week 52: number analyzed (Participants) | 275 | 553 | 286 | 540
  Change at Week 52 | -0.24 (0.69) | -0.35 (0.88) | -0.26 (0.74) | -0.41 (0.78)

34. Secondary Outcome: Change From Baseline in Number of Puffs of Daily Reliever Medication Used Per 24 Hours at Weeks 2, 4, 8, 12, 24, 36, and 52: ITT Population
Description: Participants might administered salbutamol/albuterol or levosalbutamol/levalbuterol as reliever medication as needed during the study. The number of salbutamol/albuterol or levosalbutamol/levalbuterol inhalations were recorded daily by the participants in an electronic diary/peak expiratory flow (PEF) meter. In the case that Nebulizer solutions were used as an alternative delivery method, the nebulizer dose was converted to number of puffs as per following conversion factor: salbutamol/albuterol nebulizer solution (2.5 mg) corresponds to 4 puffs.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 24, 36, and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Number of puffs of reliever medication
Arm/Group | Placebo (for Dupilumab 200 mg) q2w | Dupilumab 200 mg q2w | Placebo (for Dupilumab 300 mg) q2w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 317 | 631 | 321 | 633
Number of puffs of reliever medication
  Change at Week 2: number analyzed (Participants) | 313 | 623 | 318 | 630
  Change at Week 2 | -0.21 (1.55) | -0.56 (1.96) | -0.10 (1.71) | -0.47 (1.91)
  Change at Week 4: number analyzed (Participants) | 312 | 622 | 319 | 626
  Change at Week 4 | -0.26 (2.19) | -0.68 (2.61) | -0.34 (3.42) | -0.73 (2.42)
  Change at Week 8: number analyzed (Participants) | 308 | 617 | 314 | 607
  Change at Week 8 | -0.50 (2.23) | -1.02 (2.86) | -0.65 (2.96) | -0.94 (2.86)
  Change at Week 12: number analyzed (Participants) | 306 | 610 | 310 | 603
  Change at Week 12 | -0.52 (2.28) | -1.23 (3.03) | -0.89 (3.06) | -1.08 (2.72)
  Change at Week 24: number analyzed (Participants) | 294 | 588 | 300 | 582
  Change at Week 24 | -0.77 (2.60) | -1.27 (3.05) | -0.99 (3.21) | -1.15 (2.83)
  Change at Week 36: number analyzed (Participants) | 285 | 564 | 287 | 558
  Change at Week 36 | -0.99 (2.49) | -1.30 (2.99) | -1.06 (3.57) | -1.23 (3.01)
  Change at Week 52: number analyzed (Participants) | 270 | 522 | 265 | 521
  Change at Week 52 | -0.90 (2.58) | -1.45 (3.33) | -1.12 (3.64) | -1.39 (2.97)

35. Secondary Outcome: Change From Baseline in AQLQ (S) Self-Administered Global Score at Weeks 12, 36, and 52: ITT Population
Description: as for outcome 11
Time Frame: Baseline, Weeks 12, 36, and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo (for Dupilumab 200 mg) q2w | Dupilumab 200 mg q2w | Placebo (for Dupilumab 300 mg) q2w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 317 | 631 | 321 | 633
scores on a scale
  Change at Week 12: number analyzed (Participants) | 286 | 573 | 308 | 586
  Change at Week 12 | 0.90 (0.97) | 1.09 (1.03) | 0.94 (1.01) | 1.09 (1.09)
  Change at Week 36: number analyzed (Participants) | 271 | 554 | 295 | 548
  Change at Week 36 | 1.05 (1.08) | 1.26 (1.17) | 1.08 (1.16) | 1.33 (1.15)
  Change at Week 52: number analyzed (Participants) | 224 | 465 | 243 | 459
  Change at Week 52 | 1.00 (1.12) | 1.28 (1.16) | 1.02 (1.10) | 1.34 (1.16)

36. Secondary Outcome: Change From Baseline in European Quality of Life Working Group Health Status Measure 5 Dimensions, 5 Levels (EQ-5D-5L) Scores at Weeks 12, 24, 36, and 52: ITT Population
Description: EQ-5D-5L is a standardized health-related quality of life questionnaire developed by EuroQol Group in order to provide a simple, generic measure of health for clinical and economic appraisal. EQ-5D consists of EQ-5D descriptive system and EQ visual analogue scale (VAS). EQ-5D descriptive system comprises of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The 5D-5L systems are converted into a single index utility score between 0 to 1, where higher score indicates a better health state. EQ-5D-5L-VAS records participant's self-rated health on a vertical VAS that allows them to indicate their health state that can range from 0 (worst imaginable) to 100 (best imaginable).
Time Frame: Baseline, Weeks 12, 24, 36, and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo (for Dupilumab 200 mg) q2w | Dupilumab 200 mg q2w | Placebo (for Dupilumab 300 mg) q2w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 317 | 631 | 321 | 633
scores on a scale
  Single Index: Change at Week 12: number analyzed (Participants) | 280 | 567 | 301 | 576
  Single Index: Change at Week 12 | 0.07 (0.17) | 0.09 (0.18) | 0.08 (0.18) | 0.09 (0.18)
  Single Index: Change at Week 24: number analyzed (Participants) | 275 | 552 | 292 | 559
  Single Index: Change at Week 24 | 0.07 (0.17) | 0.09 (0.17) | 0.08 (0.18) | 0.08 (0.20)
  Single Index: Change at Week 36: number analyzed (Participants) | 264 | 548 | 290 | 537
  Single Index: Change at Week 36 | 0.08 (0.19) | 0.09 (0.20) | 0.10 (0.18) | 0.09 (0.20)
  Single Index: Change at Week 52: number analyzed (Participants) | 220 | 457 | 238 | 448
  Single Index: Change at Week 52 | 0.07 (0.20) | 0.10 (0.19) | 0.08 (0.19) | 0.10 (0.20)
  VAS Score: Change at Week 12: number analyzed (Participants) | 280 | 567 | 301 | 576
  VAS Score: Change at Week 12 | 7.69 (17.43) | 11.10 (18.90) | 6.39 (20.42) | 9.80 (19.56)
  VAS Score: Change at Week 24: number analyzed (Participants) | 275 | 552 | 292 | 559
  VAS Score: Change at Week 24 | 8.33 (17.58) | 11.44 (18.48) | 8.59 (20.37) | 9.21 (19.61)
  VAS Score: Change at Week 36: number analyzed (Participants) | 264 | 548 | 290 | 537
  VAS Score: Change at Week 36 | 9.70 (18.24) | 11.61 (19.09) | 9.31 (20.09) | 11.41 (19.40)
  VAS Score: Change at Week 52: number analyzed (Participants) | 220 | 457 | 238 | 448
  VAS Score: Change at Week 52 | 8.35 (18.51) | 12.98 (18.71) | 9.52 (20.81) | 11.90 (19.60)

37. Secondary Outcome: Change From Baseline in Hospital Anxiety and Depression Scale (HADS) Total Score at Weeks 12, 24, 36, and 52: ITT Population
Description: The HADS is a general scale to detect states of anxiety and depression already used and validated in asthma, which includes HADS-A and HADS-D subscales. The instrument is comprised of 14 items: 7 related to anxiety (HADS-A) and 7 to depression (HADS-D). Each item on the questionnaire is scored from 0-3. The anxiety/depression score is the sum of the scores of the 7 related items; one can score between 0 and 21 for either anxiety or depression. And the total score is the sum of the scores of the 14 items ranging from 0 (no symptoms) to 42 (severe symptoms), with higher scores indicating higher anxiety/depression complains.
Time Frame: Baseline, Weeks 12, 24, 36, and 52
Population: Analysis was performed on ITT population; 29 participants in Japan who received an incorrectly translated HADS questionnaire were excluded. Here 'Number analyzed' signifies number of participants with available data for specified category.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo (for Dupilumab 200 mg) q2w | Dupilumab 200 mg q2w | Placebo (for Dupilumab 300 mg) q2w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 311 | 621 | 317 | 624
scores on a scale
  Change at Week 12: number analyzed (Participants) | 274 | 551 | 297 | 569
  Change at Week 12 | -2.11 (5.29) | -1.91 (5.65) | -1.55 (6.11) | -1.98 (5.89)
  Change at Week 24: number analyzed (Participants) | 270 | 537 | 286 | 552
  Change at Week 24 | -2.17 (5.71) | -1.93 (5.97) | -1.73 (6.36) | -1.88 (6.39)
  Change at Week 36: number analyzed (Participants) | 260 | 535 | 286 | 532
  Change at Week 36 | -2.52 (5.89) | -2.02 (6.34) | -2.67 (6.80) | -2.13 (6.67)
  Change at Week 52: number analyzed (Participants) | 213 | 443 | 234 | 438
  Change at Week 52 | -2.00 (6.29) | -2.36 (6.28) | -1.86 (6.79) | -2.17 (7.04)

38. Secondary Outcome: Change From Baseline in 22-Item Sino Nasal Outcome Test (SNOT-22) Score at Weeks 12, 24, 36, and 52: ITT Population With Bilateral Nasal Polyposis/Chronic Rhinosinusitis
Description: The SNOT-22 is a validated measure of health related quality of life in sinonasal disease. It is a 22 item questionnaire with each item assigned a score ranging from 0-5. The total score may range from 0 (no disease) -110 (worst disease), lower scores represent better health related quality of life.
Time Frame: Baseline, Weeks 12, 24, 36, and 52
Population: Analysis was performed on ITT population with bilateral nasal polyposis/chronic rhinosinusitis. Here 'Number analyzed' signifies number of participants with available data for specified category.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo (for Dupilumab 200 mg) q2w | Dupilumab 200 mg q2w | Placebo (for Dupilumab 300 mg) q2w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 63 | 126 | 70 | 123
scores on a scale
  Change at Week 12: number analyzed (Participants) | 51 | 113 | 61 | 102
  Change at Week 12 | -6.82 (17.19) | -13.55 (16.85) | -11.30 (16.11) | -16.07 (20.54)
  Change at Week 24: number analyzed (Participants) | 52 | 111 | 58 | 102
  Change at Week 24 | -7.21 (17.10) | -14.68 (18.77) | -9.55 (16.04) | -17.41 (20.81)
  Change at Week 36: number analyzed (Participants) | 49 | 111 | 57 | 100
  Change at Week 36 | -6.10 (19.03) | -15.23 (18.20) | -8.51 (20.36) | -18.86 (21.34)
  Change at Week 52: number analyzed (Participants) | 42 | 89 | 49 | 85
  Change at Week 52 | -6.95 (17.10) | -15.78 (17.72) | -9.98 (18.01) | -19.81 (22.39)

39. Secondary Outcome: Change From Baseline in Standardized Rhinoconjunctivitis Quality Of Life Questionnaire, Ages 12+ (RQLQ[S]+12) Score at Weeks 12, 24, 36, and 52: ITT Population With Comorbid Allergic Rhinitis
Description: RQLQ(S)+12 is a self-administered questionnaire with standardized activities developed to measure health-related quality of life signs and symptoms that are most problematic in those 12 to 75 years of age, as a result of perennial or seasonal allergic rhinitis. There are 28 items on RQLQ(S) in 7 domains: activities (3 items), sleep (3 items), non-nose/eye symptoms (7 items), practical problems (3 items), nasal symptoms (4 items), eye symptoms (4 items) and emotional (4 items). RQLQ(S)+12 responses are based on 7-point likert scale with responses ranging from 0 (not troubled) to 6 (extremely troubled). Individual items within RQLQ(S)+12 are equally weighted. The overall score is calculated as the mean score of all items. Higher scores indicated more health-related quality of life impairment (lower scores better).
Time Frame: Baseline, Weeks 12, 24, 36, and 52
Population: Analysis was performed on ITT population with comorbid allergic rhinitis. Here 'Number analyzed' signifies number of participants with available data for specified category.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo (for Dupilumab 200 mg) q2w | Dupilumab 200 mg q2w | Placebo (for Dupilumab 300 mg) q2w | Dupilumab 300 mg q2w
Number analyzed (Participants) | 194 | 390 | 214 | 409
scores on a scale
  Change at Week 12: number analyzed (Participants) | 167 | 332 | 192 | 348
  Change at Week 12 | -0.50 (0.98) | -0.70 (0.99) | -0.44 (1.05) | -0.64 (1.06)
  Change at Week 24: number analyzed (Participants) | 164 | 322 | 182 | 342
  Change at Week 24 | -0.50 (0.92) | -0.73 (1.09) | -0.54 (1.10) | -0.60 (1.10)
  Change at Week 36: number analyzed (Participants) | 158 | 323 | 184 | 332
  Change at Week 36 | -0.56 (0.96) | -0.78 (1.15) | -0.58 (1.20) | -0.75 (1.12)
  Change at Week 52: number analyzed (Participants) | 129 | 263 | 149 | 274
  Change at Week 52 | -0.41 (0.97) | -0.90 (1.17) | -0.47 (1.33) | -0.76 (1.13)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected from signature of the informed consent form up to the final visit (Week 64) or entry in the LTS12551 open-label extension study regardless of seriousness or relationship to investigational product.
Description: Reported AEs are treatment emergent AEs that developed/worsened during 'treatment-emergent period' (from first dose of IMP until 98 days after last dose of IMP or entry in the LTS12551 study). Safety population:all participants who received at least 1 dose or part of a dose of IMP, analyzed according to treatment that participants actually received.
Groups:
- Placebo (for Dupilumab 200 mg) q2w: 2 subcutaneous injections of matched Placebo (for Dupilumab 200 mg) as a loading dose on Day 1 (Week 0), followed by a single injection q2w from Week 2 to Week 50 in combination with stable ICS and up to 2 other controller medicines (second or third controller therapy). Albuterol/salbutamol or levalbuterol/levosalbutamol was given as reliever medication. 2 participants were excluded, who were randomized to this arm but received single injection of Dupilumab 200 mg q2w and 300 mg q2w, respectively.
- Dupilumab 200 mg q2w: 2 subcutaneous injections of Dupilumab 200 mg (for a total of 400 mg) as a loading dose on Day 1 (Week 0), followed by a single 200 mg injection q2w from Week 2 to Week 50 in combination with stable ICS and up to 2 other controller medicines (second or third controller therapy). Albuterol/salbutamol or levalbuterol/levosalbutamol was given as reliever medication. 2 participants were included, who were randomized to Placebo (for Dupilumab 200 mg) arm and Dupilumab 300 mg arm, respectively but both received Dupilumab 200 mg.
- Dupilumab 300 mg q2w: 2 subcutaneous injections of Dupilumab 300 mg (for a total of 600 mg) as a loading dose on Day 1 (Week 0), followed by a single 300 mg injection q2w from Week 2 to Week 50 in combination with stable ICS and up to 2 other controller medicines (second or third controller therapy). Albuterol/salbutamol or levalbuterol/levosalbutamol was given as reliever medication. 1 participant was excluded, who was randomized to this arm but received single injection of Dupilumab 200 mg q2w. 1 participant was included, who was randomized to Placebo (for Dupilumab 200 mg) arm but received Dupilumab 300 mg.
Arm/Group | Placebo (for Dupilumab 200 mg) q2w | Dupilumab 200 mg q2w | Placebo (for Dupilumab 300 mg) q2w | Dupilumab 300 mg q2w
All-Cause Mortality (participants affected / at risk) | 3/313 | 1/631 | 0/321 | 5/632
Serious Adverse Events (participants affected / at risk) | 26/313 | 51/631 | 28/321 | 56/632
Other Adverse Events (participants affected / at risk) | 185/313 | 363/631 | 197/321 | 378/632
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (for Dupilumab 200 mg) q2w (N=313) | Dupilumab 200 mg q2w (N=631) | Placebo (for Dupilumab 300 mg) q2w (N=321) | Dupilumab 300 mg q2w (N=632)
Abscess (Infections and infestations) | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0
Atypical pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 2
Capnocytophaga infection (Infections and infestations) | 1 | 0 | 0 | 0
Chronic sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 1
Hepatitis A (Infections and infestations) | 0 | 0 | 0 | 1
Hepatitis C (Infections and infestations) | 1 | 0 | 0 | 0
Mastoiditis (Infections and infestations) | 0 | 1 | 0 | 0
Medical device site infection (Infections and infestations) | 0 | 0 | 0 | 1
Otitis media (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 4
Post procedural cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1
Pyelonephritis chronic (Infections and infestations) | 1 | 0 | 0 | 0
Tick-borne viral encephalitis (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Anaplastic thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Dysplastic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Haemangioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 1
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 0 | 1
Anaphylactic shock (Immune system disorders) | 0 | 1 | 0 | 0
Primary hyperaldosteronism (Endocrine disorders) | 1 | 0 | 0 | 0
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 1
Completed suicide (Psychiatric disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1
Major depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 1 | 1
Retinal detachment (Eye disorders) | 0 | 0 | 0 | 1
Retinal tear (Eye disorders) | 0 | 0 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 2
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 2
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0 | 1
Tachyarrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 0 | 1
Thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 10 | 11 | 5 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Eosinophilic pneumonia chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Noninfective bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diverticular perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastric volvulus (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oesophageal motility disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Strangulated umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 2
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 2
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Polychondritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Renal infarct (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1
Cervical cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Sickle cell anaemia (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 1
Impaired healing (General disorders) | 0 | 0 | 0 | 1
Injection site erythema (General disorders) | 0 | 0 | 0 | 1
Injection site inflammation (General disorders) | 0 | 0 | 0 | 1
Injection site oedema (General disorders) | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Spinal cord injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Pregnancy of partner (Social circumstances) | 0 | 1 | 0 | 0
Victim of sexual abuse (Social circumstances) | 0 | 1 | 0 | 0
Device material issue (Product Issues) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (for Dupilumab 200 mg) q2w (N=313) | Dupilumab 200 mg q2w (N=631) | Placebo (for Dupilumab 300 mg) q2w (N=321) | Dupilumab 300 mg q2w (N=632)
Bronchitis (Infections and infestations) | 47 | 73 | 43 | 70
Influenza (Infections and infestations) | 29 | 36 | 22 | 38
Sinusitis (Infections and infestations) | 27 | 36 | 29 | 26
Upper respiratory tract infection (Infections and infestations) | 37 | 70 | 48 | 77
Urinary tract infection (Infections and infestations) | 17 | 17 | 12 | 20
Viral upper respiratory tract infection (Infections and infestations) | 60 | 121 | 64 | 112
Headache (Nervous system disorders) | 26 | 47 | 25 | 40
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 16 | 21 | 15 | 18
Back pain (Musculoskeletal and connective tissue disorders) | 16 | 30 | 7 | 25
Injection site erythema (General disorders) | 13 | 76 | 22 | 98
Injection site oedema (General disorders) | 2 | 23 | 5 | 40
Accidental overdose (Injury, poisoning and procedural complications) | 16 | 31 | 16 | 34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2017-05-26): https://cdn.clinicaltrials.gov/large-docs/54/NCT02414854/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-18): https://cdn.clinicaltrials.gov/large-docs/54/NCT02414854/SAP_001.pdf